CLINICAL TRIAL: NCT02799095
Title: A Phase 1/2 Study of ALKS 4230 Administered Intravenously as Monotherapy and in Combination With Pembrolizumab in Subjects With Advanced Solid Tumors - ARTISTRY-1
Brief Title: A Study of the Effects of ALKS 4230 (Nemvaleukin Alfa) on Subjects With Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mural Oncology, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALK4230-A101
Record Dates: First submitted 2016-06-01; First posted 2016-06-14 (Estimated); Results first posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Advanced Solid Tumors
Keywords: Immunotherapy; IL-2; Interleukin-2; Solid tumors; Melanoma; Renal cell carcinoma; Non-small-cell lung cancer; Squamous cell carcinoma of the head and neck; in combination with pembrolizumab
MeSH Terms: conditions — Melanoma; Carcinoma, Renal Cell; Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ALKS 4230 (Experimental)
  Interventions: Drug: ALKS 4230
- ALKS 4230 + pembrolizumab (Experimental)
  Interventions: Drug: ALKS 4230 + pembrolizumab

INTERVENTIONS:
Drug: ALKS 4230 — Intravenous (IV) infusion over 30 minutes given daily for 5 consecutive days followed by an off-treatment period
  Arms: ALKS 4230
Drug: ALKS 4230 + pembrolizumab — IV infusion of ALKS 4230 over 30 minutes given daily for 5 consecutive days followed by an off-treatment period; pembrolizumab administered IV once with ALKS 4230 on the first day of each cycle
  Arms: ALKS 4230 + pembrolizumab

SUMMARY:
To better understand the safety and tolerability of ALKS 4230 in humans

DETAILED DESCRIPTION:
To investigate the safety and tolerability of ALKS 4230, determine the recommended Phase 2 dose (RP2D) and assess anti-tumor activity in Monotherapy and ALKS 4230 in Combination with pembrolizumab.

ELIGIBILITY:
Inclusion Criteria:

* For Part A, the subject has histological or cytological evidence of a solid tumor; for Part B, the subject has a diagnosis of melanoma or renal cell carcinoma
* All subjects must have advanced solid tumors that have returned after treatment with established approved therapies or be intolerant of established therapies
* Subjects enrolled in Part B or Part C must have at least 1 lesion that may qualify as a target lesion
* Subject can move around on their own, has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1, and has an estimated life expectancy of at least 3 months
* Subject must have adequate hematologic reserve
* Subjects must have adequate liver function
* Subjects must have adequate kidney function
* Subjects must be recovered from the effects of any prior chemotherapy, immunotherapy, other prior systemic anticancer therapy, radiotherapy or surgery
* Subjects who have received investigational agents must wait at least 4 weeks
* Females of childbearing potential must have a negative pregnancy test within 7 days of the start of treatment and on Day 1 before the first dose is administered. A female not of childbearing potential is one who has undergone bilateral oophorectomies or who is postmenopausal, defined as >45 years of age and without a menstrual period for 12 consecutive months
* Meets contraceptive requirements defined in the protocol
* Additional criteria may apply

Exclusion Criteria:

* Subject is currently pregnant or breastfeeding, or is planning to become pregnant during the study
* Subjects with an active infection or with a fever >/= 38.5 degrees C within 3 days of the first scheduled day of dosing for Cycle 1
* Subjects with active or symptomatic central nervous system metastases are excluded. Subjects with central nervous system metastases are eligible for the study if the metastases have been treated by surgery and/or radiation therapy, the subject is off corticosteroids for at least 2 weeks and the subject is neurologically stable
* Subjects have a mean QT interval corrected by the Fridericia Correction formula value of >470 msec (in females) or >450 msec (in males)
* Subjects with known hypersensitivity to any components of ALKS 4230
* Subjects with known hypersensitivity to any components of pembrolizumab (for patients in combination arm only)
* Subjects who require pharmacologic doses of corticosteroids; replacement doses, topical, ophthalmologic, and inhalational steroids are permitted
* Subjects who developed autoimmune disorders while on prior immunotherapy, including pneumonitis, nephritis, and neuropathy
* Subjects with any other concurrent uncontrolled illness, including mental illness or substance abuse, which may interfere with the ability of the subject to cooperate and participate in the study
* The subject is known to be positive for human immunodeficiency virus (HIV), hepatitis B or C, or active tuberculosis, or has a known history of tuberculosis
* Subjects with dyspnea at rest of requiring oxygen therapy
* Subjects active autoimmune disease requiring systemic treatment within the past 30 days
* Subjects who received radiotherapy within the last 4 weeks before start of study treatment administration with the exception of limited field palliative radiotherapy
* Subjects who have received systemic immunomodulatory agents within 28 days prior to C1D1.
* Subjects who have received administration of a live, attenuated vaccine within 4 weeks of Cycle 1, Day1.
* Prior solid organ and/or non-autologous hematopoietic stem cell or bone marrow transplant recipients
* Subjects who have received prior IL-2 based or IL-15 based cytokine therapy
* Additional criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2016-09-14 (Actual); Primary Completion 2023-03-27 (Actual); Study Completion 2023-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Mural Oncology
Locations (27):
- United States (12):
  - Mural Oncology Investigational Site, Denver, Colorado
  - Mural Oncology Investigational Site, Port Saint Lucie, Florida
  - Mural Oncology Investigational Site, Tampa, Florida
  - Mural Oncology Investigational Site, Lexington, Kentucky
  - Mural Oncology Investigational Site, Boston, Massachusetts
  - Mural Oncology Investigational Site, Detroit, Michigan
  - Mural Oncology Investigational Site, Buffalo, New York
  - Mural Oncology Investigational Site, New York, New York
  - Mural Oncology Investigational Site, Cleveland, Ohio
  - Mural Oncology Investigational Site, Dallas, Texas
  - Mural Oncology Investigational Site, Fairfax, Virginia
  - Mural Oncology Investigational Site, Spokane, Washington
- Australia (2):
  - Mural Oncology Investgational Site, Albury, New South Wales
  - Mural Oncology Investigational Site, Waratah, New South Wales
- Belgium (2):
  - Mural Oncology Investigational Site, Brussels, MO
  - Mural Oncology Investigational Site, Kortrijk, West-Vlaanderen
- Canada (5):
  - Mural Oncology Investigational Site, Edmonton, Alberta
  - Mural Oncology Investigational Site, Hamilton, Ontario
  - Alkermes Investigational Site, Toronto, Ontario
  - Mural Oncology Investigational Site, Montreal, Quebec
  - Mural Oncology Investigational Site, Québec, Quebec
- Mural Oncology Investigational Site, Skorzewo, Poznan, Poland
- South Korea (2):
  - Mural Oncology Investigational Site, Daejeon
  - Mural Oncology Investigational Site, Seoul
- Spain (3):
  - Mural Oncology Investigational Site, Barcelona
  - Mural Oncology Investigational Site, Madrid
  - Mural Oncology Investigational Site, Valencia

IPD SHARING:
Plan to Share IPD: No
At this time, IPD sharing has not been defined and/or decided if it will be shared.

REFERENCES:
- [Derived] Calvo E, Boni V, Dumas O, Shin SJ, Rosen SD, Chaudhry A, Debruyne PR, He X, Vaishampayan UN, McDermott DF. Nemvaleukin alfa monotherapy in patients with advanced melanoma and renal cell carcinoma: results from the phase 1/2 non-randomized ARTISTRY-1 trial. J Immunother Cancer. 2025 Aug 4;13(8):e010777. doi: 10.1136/jitc-2024-010777. PMID 40759440
- [Derived] Vaishampayan UN, Muzaffar J, Winer I, Rosen SD, Hoimes CJ, Chauhan A, Spreafico A, Lewis KD, Bruno DS, Dumas O, McDermott DF, Strauss JF, Chu QS, Gilbert L, Chaudhry A, Calvo E, Dalal R, Boni V, Ernstoff MS, Velcheti V. Nemvaleukin alfa, a modified interleukin-2 cytokine, as monotherapy and with pembrolizumab in patients with advanced solid tumors (ARTISTRY-1). J Immunother Cancer. 2024 Nov 20;12(11):e010143. doi: 10.1136/jitc-2024-010143. PMID 39567211

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 47 investigative sites in the United States, Spain, Canada, South Korea, Australia, Belgium, and Poland.
Pre-assignment Details: A total of 243 participants were enrolled in this 3-part study (Parts A, B and C) to receive nemvaleukin alfa (ALKS 4230) either as monotherapy or in combination with pembrolizumab. Selected participants (43) enrolled in Monotherapy Parts A and B, and who did not demonstrate clinical benefit were eligible to rollover to Combination Therapy Part C and were rolled over in Part C, Cohort 4.
Groups:
- Part A, Dose Escalation: Nemvaleukin Alfa 0.1 mcg/kg: Participants with advanced solid tumors received nemvaleukin alfa 0.1 microgram per kilogram (mcg/kg) intravenous (IV) infusion administration daily from Days 1 to 5 in Cycle 1 (Cycle length = 14 days) and then in Cycle 2 and subsequent cycles (each Cycle length = 21 days) until disease progression or the participant met any discontinuation criteria.
- Part A, Dose Escalation: Nemvaleukin Alfa 0.3 mcg/kg: Participants with advanced solid tumors received nemvaleukin alfa 0.3 mcg/kg IV infusion administration daily from Days 1 to 5 in Cycle 1 (Cycle length = 14 days) and then in Cycle 2 and subsequent cycles (each Cycle length = 21 days) until disease progression or the participant met any discontinuation criteria.
- Part A, Dose Escalation: Nemvaleukin Alfa 1 mcg/kg: Participants with advanced solid tumors received nemvaleukin alfa 1 mcg/kg IV infusion administration daily from Days 1 to 5 in Cycle 1 (Cycle length = 14 days) and then in Cycle 2 and subsequent cycles (each Cycle length = 21 days) until disease progression or the participant met any discontinuation criteria.
- Part A, Dose Escalation: Nemvaleukin Alfa 3 mcg/kg: Participants with advanced solid tumors received nemvaleukin alfa 3 mcg/kg IV infusion administration daily from Days 1 to 5 in Cycle 1 (Cycle length = 14 days) and then in Cycle 2 and subsequent cycles (each Cycle length = 21 days) until disease progression or the participant met any discontinuation criteria.
- Part A, Dose Escalation: Nemvaleukin Alfa 6 mcg/kg: Participants with advanced solid tumors received nemvaleukin alfa 6 mcg/kg IV infusion administration daily from Days 1 to 5 in Cycle 1 (Cycle length = 14 days) and then in Cycle 2 and subsequent cycles (each Cycle length = 21 days) until disease progression or the participant met any discontinuation criteria.
- Part A, Dose Escalation: Nemvaleukin Alfa 8 mcg/kg: Participants with advanced solid tumors received nemvaleukin alfa 8 mcg/kg IV infusion administration daily from Days 1 to 5 in Cycle 1 (Cycle length = 14 days) and then in Cycle 2 and subsequent cycles (each Cycle length = 21 days) until disease progression or the participant met any discontinuation criteria.
- Part A, Dose Escalation: Nemvaleukin Alfa 10 mcg/kg: Participants with advanced solid tumors received nemvaleukin alfa 10 mcg/kg IV infusion administration daily from Days 1 to 5 in Cycle 1 (Cycle length = 14 days) and then in Cycle 2 and subsequent cycles (each Cycle length = 21 days) until disease progression or the participant met any discontinuation criteria.
- Part B, Dose Expansion, Melanoma: Nemvaleukin Alfa 6 mcg/kg: Participants with melanoma received nemvaleukin alfa 6 mcg/kg IV infusion administration daily from Days 1 to 5 in Cycle 1 (Cycle length = 14 days) and then in Cycle 2 and subsequent cycles (each Cycle length = 21 days) until disease progression or the participant met any discontinuation criteria.
- Part B, Dose Expansion, RCC: Nemvaleukin Alfa 6 mcg/kg: Participants with renal cell carcinoma (RCC) received nemvaleukin alfa 6 mcg/kg IV infusion administration daily from Days 1 to 5 in Cycle 1 (Cycle length = 14 days) and then in Cycle 2 and subsequent cycles (each Cycle length = 21 days) until disease progression or the participant met any discontinuation criteria.
- Part C, Combination Therapy, Safety Run-in: Nemvaleukin Alfa 1 mcg/kg: Participants with any tumor type received nemvaleukin alfa 1 mcg/kg IV infusion administration daily from Days 1 to 5 in combination with pembrolizumab 200 mg IV infusion on Day 1 in each Cycle (cycle length = 21 days) for a maximum of 2 years for as long as the Participant appeared to be deriving clinical benefit (i.e., objective response or SD) and had tolerated therapy well. Participants could continue nemvaleukin alfa as monotherapy beyond the maximum of 2 years of treatment by switching to monotherapy at the joint discretion of the Investigator and Sponsor and if they did not meet any other criteria for discontinuation.
- Part C, Combination Therapy, Cohort 1 + Safety Run-in: Nemvaleukin Alfa 3mcg/kg +Pembrolizumab 200mg: Participants with programmed death receptor-1/programmed death ligand-1 (PD-1/L1) unapproved tumor types (PD-1/L1 treatment naive) received nemvaleukin alfa 3 mcg/kg IV infusion administration daily from Days 1 to 5 in combination with pembrolizumab 200 mg IV infusion on Day 1 in each Cycle (cycle length = 21 days) for a maximum of 2 years for as long as the participant appeared to be deriving clinical benefit (i.e., objective response or SD) and had tolerated therapy well. Participants could continue nemvaleukin alfa as monotherapy beyond the maximum of 2 years of treatment by switching to monotherapy at the joint discretion of the Investigator and Sponsor and if they did not meet any other criteria for discontinuation. The Safety Run-in for nemvaleukin alfa 3 mcg/kg was combined with Cohort 1 of Part C due to same dosing level and regimen.
- Part C, Combination Therapy, Cohort 2: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg: Participants with PD-1/L1 approved tumor types (PD-1/L1 treatment pretreated) received nemvaleukin alfa 3 mcg/kg IV infusion administration daily from Days 1 to 5 in combination with pembrolizumab 200 mg IV infusion on Day 1 in each Cycle (cycle length = 21 days) for a maximum of 2 years for as long as the participant appeared to be deriving clinical benefit (i.e., objective response or SD) and had tolerated therapy well. Participants could continue nemvaleukin alfa as monotherapy beyond the maximum of 2 years of treatment by switching to monotherapy at the joint discretion of the Investigator and Sponsor and if they did not meet any other criteria for discontinuation.
- Part C, Combination Therapy, Cohort 3: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg: Participants with PD-1/L1 approved tumor types (PD-1/L1 treatment naive) received nemvaleukin alfa 3 mcg/kg IV infusion administration daily from Days 1 to 5 in combination with pembrolizumab 200 mg IV infusion on Day 1 in each Cycle (cycle length = 21 days) for a maximum of 2 years for as long as the participant appeared to be deriving clinical benefit (i.e., objective response or SD) and had tolerated therapy well. Participants could continue nemvaleukin alfa as monotherapy beyond the maximum of 2 years of treatment by switching to monotherapy at the joint discretion of the Investigator and Sponsor and if they did not meet any other criteria for discontinuation.
- Part C, Combination Therapy, Rollover, Cohort 4: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg: Participants rolled over from Parts A or B received nemvaleukin alfa 3 mcg/kg IV infusion administration daily from Days 1 to 5 in combination with pembrolizumab 200 mg IV infusion on Day 1 in each Cycle (cycle length = 21 days) for a maximum of 2 years for as long as the participant appeared to be deriving clinical benefit (i.e., objective response or SD) and had tolerated therapy well. Participants could continue nemvaleukin alfa as monotherapy beyond the maximum of 2 years of treatment by switching to monotherapy at the joint discretion of the Investigator and Sponsor and if they did not meet any other criteria for discontinuation.
- Part C, Combination Therapy, Cohort 5: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg: Participants with melanoma received nemvaleukin alfa 6 mcg/kg IV infusion administration daily from Days 1 to 5 in combination with pembrolizumab 200 mg IV infusion on Day 1 in each Cycle (cycle length = 21 days) for a maximum of 2 years for as long as the participant appeared to be deriving clinical benefit (i.e., objective response or SD) and had tolerated therapy well. Participants could continue nemvaleukin alfa as monotherapy beyond the maximum of 2 years of treatment by switching to monotherapy at the joint discretion of the Investigator and Sponsor and if they did not meet any other criteria for discontinuation.
- Part C, Combination Therapy, Cohort 6: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg: Participants with non-small-cell lung cancer (NSCLC) received nemvaleukin alfa 6 mcg/kg IV infusion administration daily from Days 1 to 5 in combination with pembrolizumab 200 mg IV infusion on Day 1 in each Cycle (cycle length = 21 days) for a maximum of 2 years for as long as the participant appeared to be deriving clinical benefit (i.e., objective response or SD) and had tolerated therapy well. Participants could continue nemvaleukin alfa as monotherapy beyond the maximum of 2 years of treatment by switching to monotherapy at the joint discretion of the Investigator and Sponsor and if they did not meet any other criteria for discontinuation.
- Part C, Combination Therapy, Cohort 7: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg: Participants with squamous cell carcinoma of the head and neck (SCCHN) received nemvaleukin alfa 6 mcg/kg IV infusion administration daily from Days 1 to 5 in combination with pembrolizumab 200 mg IV infusion on Day 1 in each Cycle (cycle length = 21 days) for a maximum of 2 years for as long as the participant appeared to be deriving clinical benefit (i.e., objective response or SD) and had tolerated therapy well. Participants could continue nemvaleukin alfa as monotherapy beyond the maximum of 2 years of treatment by switching to monotherapy at the joint discretion of the Investigator and Sponsor and if they did not meet any other criteria for discontinuation.
Period: Part A
Arm/Group | Part A, Dose Escalation: Nemvaleukin Alfa 0.1 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 0.3 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 1 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 3 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 6 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 8 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 10 mcg/kg | Part B, Dose Expansion, Melanoma: Nemvaleukin Alfa 6 mcg/kg | Part B, Dose Expansion, RCC: Nemvaleukin Alfa 6 mcg/kg | Part C, Combination Therapy, Safety Run-in: Nemvaleukin Alfa 1 mcg/kg | Part C, Combination Therapy, Cohort 1 + Safety Run-in: Nemvaleukin Alfa 3mcg/kg +Pembrolizumab 200mg | Part C, Combination Therapy, Cohort 2: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 3: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Rollover, Cohort 4: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 5: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 6: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 7: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg
Started | 5 | 4 | 7 | 8 | 12 | 3 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 5 | 4 | 7 | 8 | 12 | 3 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 1 | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Progressive Disease | 3 | 3 | 3 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Clinical Progression | 1 | 0 | 2 | 1 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Deviation | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Rolled Over to Part C, Cohort 4 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B
Arm/Group | Part A, Dose Escalation: Nemvaleukin Alfa 0.1 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 0.3 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 1 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 3 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 6 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 8 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 10 mcg/kg | Part B, Dose Expansion, Melanoma: Nemvaleukin Alfa 6 mcg/kg | Part B, Dose Expansion, RCC: Nemvaleukin Alfa 6 mcg/kg | Part C, Combination Therapy, Safety Run-in: Nemvaleukin Alfa 1 mcg/kg | Part C, Combination Therapy, Cohort 1 + Safety Run-in: Nemvaleukin Alfa 3mcg/kg +Pembrolizumab 200mg | Part C, Combination Therapy, Cohort 2: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 3: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Rollover, Cohort 4: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 5: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 6: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 7: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 47 (Participants who were assigned in Part B to receive specified treatment.) | 27 (Participants who were assigned in Part B to receive specified treatment.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 44 | 26 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Progressive Disease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Rolled Over to Part C, Cohort 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 26 | 12 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part C
Arm/Group | Part A, Dose Escalation: Nemvaleukin Alfa 0.1 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 0.3 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 1 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 3 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 6 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 8 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 10 mcg/kg | Part B, Dose Expansion, Melanoma: Nemvaleukin Alfa 6 mcg/kg | Part B, Dose Expansion, RCC: Nemvaleukin Alfa 6 mcg/kg | Part C, Combination Therapy, Safety Run-in: Nemvaleukin Alfa 1 mcg/kg | Part C, Combination Therapy, Cohort 1 + Safety Run-in: Nemvaleukin Alfa 3mcg/kg +Pembrolizumab 200mg | Part C, Combination Therapy, Cohort 2: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 3: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Rollover, Cohort 4: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 5: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 6: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 7: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 (Participants who were assigned in Part C to receive specified treatment.) | 42 (Participants who were assigned in Part C to receive specified treatment.) | 26 (Participants who were assigned in Part C to receive specified treatment.) | 26 (Participants who were assigned in Part C to receive specified treatment.) | 43 (Participants were rolled over from Monotherapy (Part A or B).) | 3 (Participants who were assigned in Part C to receive specified treatment.) | 21 (Participants who were assigned in Part C to receive specified treatment.) | 2 (Participants who were assigned in Part C to receive specified treatment.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 8 | 2 | 1 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 41 | 26 | 22 | 35 | 1 | 20 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 5 | 6 | 8 | 1 | 8 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 3 | 0 | 0 | 0
Not completed — Progressive Disease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 13 | 2 | 0 | 1 | 0 | 0 | 0
Not completed — Clinical Progression | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 15 | 13 | 21 | 0 | 12 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least 1 dose of nemvaleukin alfa or pembrolizumab. Selected participants (43) enrolled in Monotherapy Parts A and B, and who did not demonstrate clinical benefit were eligible to rollover to Combination Therapy Part C and were rolled over in Part C, Cohort 4.
Groups:
- Part A, Dose Escalation: Nemvaleukin Alfa 0.1 mcg/kg: Participants with advanced solid tumors received nemvaleukin alfa 0.1 mcg/kg IV infusion administration daily from Days 1 to 5 in Cycle 1 (Cycle length = 14 days) and then in Cycle 2 and subsequent cycles (each Cycle length = 21 days) until disease progression or the participant met any discontinuation criteria.
- Part B, Dose Expansion, RCC: Nemvaleukin 6 Alfa mcg/kg: Participants with RCC received nemvaleukin alfa 6 mcg/kg IV infusion administration daily from Days 1 to 5 in Cycle 1 (Cycle length = 14 days) and then in Cycle 2 and subsequent cycles (each Cycle length = 21 days) until disease progression or the participant met any discontinuation criteria.
- Part C, Combination Therapy, Cohort 1 + Safety Run-in: Nemvaleukin Alfa 3mcg/kg +Pembrolizumab 200mg: Participants with PD-1/L1 unapproved tumor types (PD-1/L1 treatment naive) received nemvaleukin alfa 3 mcg/kg IV infusion administration daily from Days 1 to 5 in combination with pembrolizumab 200 mg IV infusion on Day 1 in each Cycle (cycle length = 21 days) for a maximum of 2 years for as long as the participant appeared to be deriving clinical benefit (i.e., objective response or SD) and had tolerated therapy well. Participants could continue nemvaleukin alfa as monotherapy beyond the maximum of 2 years of treatment by switching to monotherapy at the joint discretion of the Investigator and Sponsor and if they did not meet any other criteria for discontinuation. The Safety Run-in for nemvaleukin alfa 3 mcg/kg was combined with Cohort 1 of Part C due to same dosing level and regimen.
- Part C, Combination Therapy, Rollover, Cohort 4: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg: Participants rollover from Parts A or B received nemvaleukin alfa 3 mcg/kg IV infusion administration daily from Days 1 to 5 in combination with pembrolizumab 200 mg IV infusion on Day 1 in each Cycle (cycle length = 21 days) for a maximum of 2 years for as long as the participant appeared to be deriving clinical benefit (i.e., objective response or SD) and had tolerated therapy well. Participants could continue nemvaleukin alfa as monotherapy beyond the maximum of 2 years of treatment by switching to monotherapy at the joint discretion of the Investigator and Sponsor and if they did not meet any other criteria for discontinuation.
- Part C, Combination Therapy, Cohort 6: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg: Participants with NSCLC received nemvaleukin alfa 6 mcg/kg IV infusion administration daily from Days 1 to 5 in combination with pembrolizumab 200 mg IV infusion on Day 1 in each Cycle (cycle length = 21 days) for a maximum of 2 years for as long as the participant appeared to be deriving clinical benefit (i.e., objective response or SD) and had tolerated therapy well. Participants could continue nemvaleukin alfa as monotherapy beyond the maximum of 2 years of treatment by switching to monotherapy at the joint discretion of the Investigator and Sponsor and if they did not meet any other criteria for discontinuation.
- Part C, Combination Therapy, Cohort 7: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg: Participants with SCCHN received nemvaleukin alfa 6 mcg/kg IV infusion administration daily from Days 1 to 5 in combination with pembrolizumab 200 mg IV infusion on Day 1 in each Cycle (cycle length = 21 days) for a maximum of 2 years for as long as the participant appeared to be deriving clinical benefit (i.e., objective response or SD) and had tolerated therapy well. Participants could continue nemvaleukin alfa as monotherapy beyond the maximum of 2 years of treatment by switching to monotherapy at the joint discretion of the Investigator and Sponsor and if they did not meet any other criteria for discontinuation.
- Total: Total of all reporting groups
Arm/Group | Part A, Dose Escalation: Nemvaleukin Alfa 0.1 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 0.3 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 1 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 3 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 6 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 8 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 10 mcg/kg | Part B, Dose Expansion, Melanoma: Nemvaleukin Alfa 6 mcg/kg | Part B, Dose Expansion, RCC: Nemvaleukin 6 Alfa mcg/kg | Part C, Combination Therapy, Safety Run-in: Nemvaleukin Alfa 1 mcg/kg | Part C, Combination Therapy, Cohort 1 + Safety Run-in: Nemvaleukin Alfa 3mcg/kg +Pembrolizumab 200mg | Part C, Combination Therapy, Cohort 2: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 3: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Rollover, Cohort 4: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 5: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 6: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 7: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg | Total
Number analyzed (Participants) | 5 | 4 | 7 | 8 | 12 | 3 | 7 | 47 | 27 | 3 | 42 | 26 | 26 | 43 | 3 | 21 | 2 | 286
Age, Customized [Count of Participants; unit: Participants] — Population: Here, "Number Analyzed" signifies participants who were evaluable for specified parts.
  Participants
    Part A: number analyzed (Participants) | 5 | 4 | 7 | 8 | 12 | 3 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 46
    Part A: 18 to 64 years | 5 | 3 | 5 | 4 | 4 | 3 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 28
    Part A: 65 to 84 years | 0 | 1 | 2 | 4 | 8 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 18
    Part A: > 84 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Part B: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 47 | 27 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 74
    Part B: 18 to 64 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 20 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 30
    Part B: 65 to 84 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 27 | 17 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 44
    Part B: > 84 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  | 0
    Part C: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 42 | 26 | 26 | 43 | 3 | 21 | 2 | 166
    Part C: 18 to 64 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 30 | 20 | 15 | 18 | 1 | 11 | 1 | 96
    Part C: 65 to 84 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 12 | 6 | 11 | 25 | 2 | 9 | 1 | 69
    Part C: > 84 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Here, "Number Analyzed" signifies participants who were evaluable for specified parts.
  Participants
    Part A: number analyzed (Participants) | 5 | 4 | 7 | 8 | 12 | 3 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 46
    Part A: Female | 1 | 1 | 0 | 4 | 7 | 2 | 4 |  |  |  |  |  |  |  |  |  |  | 19
    Part A: Male | 4 | 3 | 7 | 4 | 5 | 1 | 3 |  |  |  |  |  |  |  |  |  |  | 27
    Part B: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 47 | 27 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 74
    Part B: Female |  |  |  |  |  |  |  | 22 | 3 |  |  |  |  |  |  |  |  | 25
    Part B: Male |  |  |  |  |  |  |  | 25 | 24 |  |  |  |  |  |  |  |  | 49
    Part C: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 42 | 26 | 26 | 43 | 3 | 21 | 2 | 166
    Part C: Female |  |  |  |  |  |  |  |  |  | 1 | 28 | 12 | 13 | 18 | 1 | 7 | 1 | 81
    Part C: Male |  |  |  |  |  |  |  |  |  | 2 | 14 | 14 | 13 | 25 | 2 | 14 | 1 | 85
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Here, "Number Analyzed" signifies participants who were evaluable for specified parts.
  Participants
    Part A: number analyzed (Participants) | 5 | 4 | 7 | 8 | 12 | 3 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 46
    Part A: Hispanic or Latino | 1 | 0 | 0 | 0 | 0 | 0 | 1 |  |  |  |  |  |  |  |  |  |  | 2
    Part A: Not Hispanic or Latino | 4 | 4 | 7 | 8 | 12 | 3 | 6 |  |  |  |  |  |  |  |  |  |  | 44
    Part A: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |  |  |  |  |  |  |  | 0
    Part B: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 47 | 27 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 74
    Part B: Hispanic or Latino |  |  |  |  |  |  |  | 0 | 1 |  |  |  |  |  |  |  |  | 1
    Part B: Not Hispanic or Latino |  |  |  |  |  |  |  | 47 | 26 |  |  |  |  |  |  |  |  | 73
    Part B: Unknown or Not Reported |  |  |  |  |  |  |  | 0 | 0 |  |  |  |  |  |  |  |  | 0
    Part C: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 42 | 26 | 26 | 43 | 3 | 21 | 2 | 166
    Part C: Hispanic or Latino |  |  |  |  |  |  |  |  |  | 0 | 1 | 1 | 2 | 1 | 0 | 1 | 0 | 6
    Part C: Not Hispanic or Latino |  |  |  |  |  |  |  |  |  | 3 | 40 | 25 | 24 | 42 | 3 | 20 | 2 | 159
    Part C: Unknown or Not Reported |  |  |  |  |  |  |  |  |  | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Here, "Number Analyzed" signifies participants who were evaluable for specified parts.
  Participants
    Part A: number analyzed (Participants) | 5 | 4 | 7 | 8 | 12 | 3 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 46
    Part A: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |  |  |  |  |  |  |  | 0
    Part A: Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |  |  |  |  |  |  |  | 0
    Part A: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |  |  |  |  |  |  |  | 0
    Part A: Black or African American | 0 | 0 | 1 | 0 | 2 | 1 | 0 |  |  |  |  |  |  |  |  |  |  | 4
    Part A: White | 5 | 4 | 6 | 8 | 10 | 2 | 6 |  |  |  |  |  |  |  |  |  |  | 41
    Part A: More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  |  |  |  |  |  |  |  | 0
    Part A: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 1 |  |  |  |  |  |  |  |  |  |  | 1
    Part B: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 47 | 27 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 74
    Part B: American Indian or Alaska Native |  |  |  |  |  |  |  | 0 | 0 |  |  |  |  |  |  |  |  | 0
    Part B: Asian |  |  |  |  |  |  |  | 5 | 1 |  |  |  |  |  |  |  |  | 6
    Part B: Native Hawaiian or Other Pacific Islander |  |  |  |  |  |  |  | 0 | 0 |  |  |  |  |  |  |  |  | 0
    Part B: Black or African American |  |  |  |  |  |  |  | 0 | 1 |  |  |  |  |  |  |  |  | 1
    Part B: White |  |  |  |  |  |  |  | 42 | 25 |  |  |  |  |  |  |  |  | 67
    Part B: More than one race |  |  |  |  |  |  |  | 0 | 0 |  |  |  |  |  |  |  |  | 0
    Part B: Unknown or Not Reported |  |  |  |  |  |  |  | 0 | 0 |  |  |  |  |  |  |  |  | 0
    Part C: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 42 | 26 | 26 | 43 | 3 | 21 | 2 | 166
    Part C: American Indian or Alaska Native |  |  |  |  |  |  |  |  |  | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Part C: Asian |  |  |  |  |  |  |  |  |  | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 3
    Part C: Native Hawaiian or Other Pacific Islander |  |  |  |  |  |  |  |  |  | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Part C: Black or African American |  |  |  |  |  |  |  |  |  | 0 | 7 | 3 | 3 | 1 | 0 | 1 | 0 | 15
    Part C: White |  |  |  |  |  |  |  |  |  | 3 | 34 | 20 | 22 | 40 | 3 | 18 | 2 | 142
    Part C: More than one race |  |  |  |  |  |  |  |  |  | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Part C: Unknown or Not Reported |  |  |  |  |  |  |  |  |  | 0 | 1 | 2 | 1 | 1 | 0 | 1 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: Part A: Number of Participants With Dose-limiting Toxicities (DLTs) Based on Common Terminology Criteria for Adverse Events (CTCAE)
Description: DLT was defined by any of following events possibly, probably, or definitely related to ALKS 4230: Grade 4 neutrophil count decreased (neutropenia); Febrile neutropenia; CTCAE Grade 4 thrombocytopenia; Thrombocytopenia; Any Grade 3 cardiac or central nervous system toxicity; Liver transaminase elevation higher than 8*upper limit of normal (ULN) or total bilirubin higher than 6*ULN; Grade 4 hypoalbuminemia; Fever more than (>) 40 degree Celsius (°C) sustained for >24 hours; Hypotension required the use of pressors or prolonged hospitalization (>48 hours) for hypotension requiring medical intervention; Grade 3 or higher electrolyte abnormalities; Increase in amylase or lipase; Grade 3 or higher nausea, vomiting, or diarrhea; Any other Grade 4 nonhematologic toxicity or any other Grade 3 non-hematologic toxicity; Any other toxicity or adverse event (AE) not defined above that resulted in participant removal from the study or discontinuation of dosing by the Investigator.
Time Frame: Cycle 1 Day 1 through Cycle 2 Day 15 (Cycle 1 length = 14 days; Cycle 2 length= 21 days)
Population: Safety population included all participants who received at least 1 dose of nemvaleukin alfa or pembrolizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Dose Escalation: Nemvaleukin Alfa 0.1 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 0.3 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 1 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 3 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 6 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 8 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 10 mcg/kg
Number analyzed (Participants) | 5 | 4 | 7 | 8 | 12 | 3 | 7
Participants | 0 | 0 | 0 | 2 | 3 | 0 | 1

2. Primary Outcome: Parts A, B, and C: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: TEAEs were defined as AEs that were newly occurring or worsening from the time of the first dose of study drug. An AE was any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product.
Time Frame: From first dose of study drug until 30 days after last dose (up to 10 months for Part A; up to 41.3 months for Part B; up to 51.5 months for Part C)
Population: Safety population included all participants who received at least 1 dose of nemvaleukin alfa or pembrolizumab.
Measure: Count of Participants; unit: Participants
Groups:
- Part B, Dose Expansion, RCC: Nemvaleukin Alfa 6 mcg/kg: Participants with RCC received nemvaleukin alfa 6 mcg/kg IV infusion administration daily from Days 1 to 5 in Cycle 1 (Cycle length = 14 days) and then in Cycle 2 and subsequent cycles (each Cycle length = 21 days) until disease progression or the participant met any discontinuation criteria.
- Part C, Combination Therapy, Cohort 1 +Safety Run-in: Nemvaleukin Alfa 3 mcg/kg+Pembrolizumab 200 mg: Participants with PD-1/L1 unapproved tumor types (PD-1/L1 treatment naive) received nemvaleukin alfa 3 mcg/kg IV infusion administration daily from Days 1 to 5 in combination with pembrolizumab 200 mg IV infusion on Day 1 in each Cycle (cycle length = 21 days) for a maximum of 2 years for as long as the participant appeared to be deriving clinical benefit (i.e., objective response or SD) and had tolerated therapy well. Participants could continue nemvaleukin alfa as monotherapy beyond the maximum of 2 years of treatment by switching to monotherapy at the joint discretion of the Investigator and Sponsor and if they did not meet any other criteria for discontinuation. The Safety Run-in for nemvaleukin alfa 3 mcg/kg was combined with Cohort 1 of Part C due to same dosing level and regimen.
- Part C, Combination Therapy, Cohort 5: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg: Participants with melanoma received nemvaleukin alfa 6 mcg/kg IV administration daily from Days 1 to 5 in combination with pembrolizumab 200 mg IV infusion on Day 1 in each Cycle (cycle length = 21 days) for a maximum of 2 years for as long as the participant appeared to be deriving clinical benefit (i.e., objective response or SD) and had tolerated therapy well. Participants could continue nemvaleukin alfa as monotherapy beyond the maximum of 2 years of treatment by switching to monotherapy at the joint discretion of the Investigator and Sponsor and if they did not meet any other criteria for discontinuation.
Arm/Group | Part A, Dose Escalation: Nemvaleukin Alfa 0.1 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 0.3 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 1 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 3 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 6 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 8 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 10 mcg/kg | Part B, Dose Expansion, Melanoma: Nemvaleukin Alfa 6 mcg/kg | Part B, Dose Expansion, RCC: Nemvaleukin Alfa 6 mcg/kg | Part C, Combination Therapy, Safety Run-in: Nemvaleukin Alfa 1 mcg/kg | Part C, Combination Therapy, Cohort 1 +Safety Run-in: Nemvaleukin Alfa 3 mcg/kg+Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 2: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 3: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Rollover, Cohort 4: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 5: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 6: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 7: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg
Number analyzed (Participants) | 5 | 4 | 7 | 8 | 12 | 3 | 7 | 47 | 27 | 3 | 42 | 26 | 26 | 43 | 3 | 21 | 2
Participants | 5 | 4 | 7 | 8 | 12 | 3 | 7 | 46 | 27 | 3 | 42 | 26 | 26 | 39 | 3 | 21 | 2

3. Primary Outcome: Parts A, B, and C: Number of Participants With TEAEs by Severity Grading
Description: TEAEs were defined as AEs that were newly occurring or worsening from the time of the first dose of study drug. Severity was graded according to the National Cancer Institute (NCI) CTCAE (version 4.03) where, Grade 1: Mild- asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2: Moderate- minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living (ADL) Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL. Grade 4: Life-threatening consequences; urgent intervention indicated. Grade 5: Death related to AE. As planned, Grades 1 and 2 were combined for reporting.
Time Frame: as for outcome 2
Population: Safety population included all participants who received at least 1 dose of nemvaleukin alfa or pembrolizumab.
Measure: Count of Participants; unit: Participants
Groups:
- Part C, Combination Therapy, Safety Run-in: Nemvaleukin Alfa 1 mcg/kg: Participants with any tumor type received nemvaleukin alfa 1 mcg/kg IV infusion administration daily from Days 1 to 5 in combination with pembrolizumab 200 mg IV infusion on Day 1 in each Cycle (cycle length = 21 days) for a maximum of 2 years for as long as the Participant appeared to be deriving clinical benefit (i.e., objective response or SD) and had tolerated therapy well. Participants could continue nemvaleukin as monotherapy beyond the maximum of 2 years of treatment by switching to monotherapy at the joint discretion of the Investigator and Sponsor and if they did not meet any other criteria for discontinuation.
- Part C, Combination Therapy, Cohort 1 +Safety Run-in: Nemvaleukin Alfa 3 mcg/kg +Pembrolizumab 200mg: Participants with PD-1/L1 unapproved tumor types (PD-1/L1 treatment naive) received nemvaleukin 3 mcg/kg IV infusion administration daily from Days 1 to 5 in combination with pembrolizumab 200 mg IV infusion on Day 1 in each Cycle (cycle length = 21 days) for a maximum of 2 years for as long as the participant appeared to be deriving clinical benefit (i.e., objective response or SD) and had tolerated therapy well. Participants could continue nemvaleukin as monotherapy beyond the maximum of 2 years of treatment by switching to monotherapy at the joint discretion of the Investigator and Sponsor and if they did not meet any other criteria for discontinuation. The Safety Run-in for nemvaleukin 3 mcg/kg was combined with Cohort 1 of Part C due to same dosing level and regimen.
- Part C, Combination Therapy, Cohort 2: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg: Participants with PD-1/L1 approved tumor types (PD-1/L1 treatment pretreated) received nemvaleukin alfa 3 mcg/kg IV infusion administration daily from Days 1 to 5 in combination with pembrolizumab 200 mg IV infusion on Day 1 in each Cycle (cycle length = 21 days) for a maximum of 2 years for as long as the participant appeared to be deriving clinical benefit (i.e., objective response or SD) and had tolerated therapy well. Participants could continue nemvaleukin as monotherapy beyond the maximum of 2 years of treatment by switching to monotherapy at the joint discretion of the Investigator and Sponsor and if they did not meet any other criteria for discontinuation.
Arm/Group | Part A, Dose Escalation: Nemvaleukin Alfa 0.1 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 0.3 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 1 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 3 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 6 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 8 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 10 mcg/kg | Part B, Dose Expansion, Melanoma: Nemvaleukin Alfa 6 mcg/kg | Part B, Dose Expansion, RCC: Nemvaleukin Alfa 6 mcg/kg | Part C, Combination Therapy, Safety Run-in: Nemvaleukin Alfa 1 mcg/kg | Part C, Combination Therapy, Cohort 1 +Safety Run-in: Nemvaleukin Alfa 3 mcg/kg +Pembrolizumab 200mg | Part C, Combination Therapy, Cohort 2: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 3: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Rollover, Cohort 4: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 5: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 6: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 7: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg
Number analyzed (Participants) | 5 | 4 | 7 | 8 | 12 | 3 | 7 | 47 | 27 | 3 | 42 | 26 | 26 | 43 | 3 | 21 | 2
Participants
  Participants With Grade 1 and 2 TEAEs | 2 | 3 | 4 | 2 | 3 | 1 | 1 | 6 | 5 | 3 | 16 | 7 | 6 | 13 | 1 | 4 | 0
  Participants With Grade 3 TEAEs | 3 | 1 | 3 | 6 | 8 | 2 | 3 | 28 | 16 | 0 | 19 | 14 | 15 | 21 | 1 | 16 | 1
  Participants With Grade 4 TEAEs | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 12 | 5 | 0 | 4 | 5 | 5 | 4 | 1 | 1 | 1
  Participants With Grade 5 TEAEs | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 0

4. Primary Outcome: Parts B and C: Overall Response Rate (ORR) Based on Response Evaluation Criteria in Solid Tumors (RECIST) Version (v) 1.1
Description: ORR rate was defined as the percentage of participants with objective evidence of CR or PR based on RECIST v1.1. Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<) 10 millimeters (mm). Partial Response (PR): At least a 30 percent (%) decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From first dose of study drug up to 40.3 months for Part B and up to 50.5 months for Part C
Population: The antitumor evaluable population consisted of participants who complete 2 cycles of therapy and had at least one follow-up scan.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Part C, Combination Therapy, Cohort 1 +Safety Run-in: Nemvaleukin Alfa 3 mcg/kg +Pembrolizumab 200mg: Participants with PD-1/L1 unapproved tumor types (PD-1/L1 treatment naive) received nemvaleukin alfa 3 mcg/kg IV infusion administration daily from Days 1 to 5 in combination with pembrolizumab 200 mg IV infusion on Day 1 in each Cycle (cycle length = 21 days) for a maximum of 2 years for as long as the participant appeared to be deriving clinical benefit (i.e., objective response or SD) and had tolerated therapy well. Participants could continue nemvaleukin alfa as monotherapy beyond the maximum of 2 years of treatment by switching to monotherapy at the joint discretion of the Investigator and Sponsor and if they did not meet any other criteria for discontinuation. The Safety Run-in for nemvaleukin alfa 3 mcg/kg was combined with Cohort 1 of Part C due to same dosing level and regimen.
Arm/Group | Part B, Dose Expansion, Melanoma: Nemvaleukin Alfa 6 mcg/kg | Part B, Dose Expansion, RCC: Nemvaleukin Alfa 6 mcg/kg | Part C, Combination Therapy, Safety Run-in: Nemvaleukin Alfa 1 mcg/kg | Part C, Combination Therapy, Cohort 1 +Safety Run-in: Nemvaleukin Alfa 3 mcg/kg +Pembrolizumab 200mg | Part C, Combination Therapy, Cohort 2: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 3: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Rollover, Cohort 4: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 5: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 6: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 7: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg
Number analyzed (Participants) | 46 | 22 | 3 | 36 | 22 | 21 | 39 | 3 | 18 | 2
percentage of participants | 8.7 [2.4 to 20.8] | 13.6 [2.9 to 34.9] | 0.0 [0.0 to 70.8] | 13.9 [4.7 to 29.5] | 0.0 [0.0 to 15.4] | 28.6 [11.3 to 52.2] | 7.7 [1.6 to 20.9] | 66.7 [9.4 to 99.2] | 11.1 [1.4 to 34.7] | 50.0 [1.3 to 98.7]

5. Secondary Outcome: Parts A, B, and C: Serum Concentrations of Nemvaleukin Alfa
Description: Cycle 1 length = 14 days for Part A and 21 days for Part B and C; Cycle 2 length= 21 days for all parts.
Time Frame: Cycle 1 and 2 Day 1: 0, 0.5, 1, 2, 4, 8, 16, and 24 hours post-dose; Cycle 1 Day 5: 0, 0.5, 1, 2, 4, 8, 16, 24, and 72 hours post-dose; Cycle 2 Day 5: 0, 0.5, 1, 2, 4, 8, 16, 24, 72, and 240 hours post-dose
Population: The pharmacokinetic (PK) population consisted of all participants who received at least 1 dose of nemvaleukin alfa and had at least 1 measurable serum concentration of nemvaleukin alfa at any scheduled PK time point. Here, "overall number of participants analyzed" signifies participants who were evaluable for this outcome measure and "number analyzed" signifies participants who were evaluable at specified timepoints.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Groups:
- Part C, Combination Therapy, Safety Run-in: Nemvaleukin Alfa 3 mcg/kg: Participants with PD-1/L1 unapproved tumor types (PD-1/L1 treatment naive) received nemvaleukin alfa 3 mcg/kg IV infusion administration daily from Days 1 to 5 in combination with pembrolizumab 200 mg IV infusion on Day 1 in each Cycle (cycle length = 21 days) for a maximum of 2 years for as long as the Participant appeared to be deriving clinical benefit (i.e., objective response or SD) and had tolerated therapy well. Participants could continue nemvaleukin alfa as monotherapy beyond the maximum of 2 years of treatment by switching to monotherapy at the joint discretion of the Investigator and Sponsor and if they did not meet any other criteria for discontinuation.
- Part C, Combination Therapy, Cohort 1: Nemvaleukin Alfa 3 mcg/kg +Pembrolizumab 200mg: Participants with PD-1/L1 unapproved tumor types (PD-1/L1 treatment naive) received nemvaleukin alfa 3 mcg/kg infusion IV administration daily from Days 1 to 5 in combination with pembrolizumab 200 mg IV infusion on Day 1 in each Cycle (cycle length = 21 days) for a maximum of 2 years for as long as the participant appeared to be deriving clinical benefit (i.e., objective response or SD) and had tolerated therapy well. Participants could continue nemvaleukin alfa as monotherapy beyond the maximum of 2 years of treatment by switching to monotherapy at the joint discretion of the Investigator and Sponsor and if they did not meet any other criteria for discontinuation.
- Part C, Combination Therapy, Cohort 7: Nemvaleukin 6 Alfa mcg/kg + Pembrolizumab 200 mg: Participants with SCCHN received nemvaleukin alfa 6 mcg/kg IV infusion administration daily from Days 1 to 5 in combination with pembrolizumab 200 mg IV infusion on Day 1 in each Cycle (cycle length = 21 days) for a maximum of 2 years for as long as the participant appeared to be deriving clinical benefit (i.e., objective response or SD) and had tolerated therapy well. Participants could continue nemvaleukin alfa as monotherapy beyond the maximum of 2 years of treatment by switching to monotherapy at the joint discretion of the Investigator and Sponsor and if they did not meet any other criteria for discontinuation.
Arm/Group | Part A, Dose Escalation: Nemvaleukin Alfa 0.1 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 0.3 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 1 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 3 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 6 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 8 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 10 mcg/kg | Part B, Dose Expansion, Melanoma: Nemvaleukin Alfa 6 mcg/kg | Part B, Dose Expansion, RCC: Nemvaleukin Alfa 6 mcg/kg | Part C, Combination Therapy, Safety Run-in: Nemvaleukin Alfa 1 mcg/kg | Part C, Combination Therapy, Safety Run-in: Nemvaleukin Alfa 3 mcg/kg | Part C, Combination Therapy, Cohort 1: Nemvaleukin Alfa 3 mcg/kg +Pembrolizumab 200mg | Part C, Combination Therapy, Cohort 2: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 3: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Rollover, Cohort 4: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 5: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 6: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 7: Nemvaleukin 6 Alfa mcg/kg + Pembrolizumab 200 mg
Number analyzed (Participants) | 5 | 4 | 7 | 8 | 12 | 3 | 7 | 45 | 27 | 3 | 6 | 35 | 25 | 26 | 43 | 3 | 20 | 2
nanograms per milliliter (ng/mL)
  Cycle 1 Day 1: 0 hour: number analyzed (Participants) | 5 | 4 | 7 | 8 | 11 | 3 | 7 | 45 | 27 | 3 | 6 | 35 | 25 | 26 | 43 | 3 | 19 | 2
  Cycle 1 Day 1: 0 hour | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.0137 (0.0917) | 0.0329 (0.171) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.0151 (0.0988) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)
  Cycle 1 Day 1: 0.5 hour: number analyzed (Participants) | 5 | 3 | 5 | 6 | 9 | 3 | 5 | 41 | 26 | 2 | 6 | 29 | 23 | 25 | 33 | 2 | 15 | 2
  Cycle 1 Day 1: 0.5 hour | 2.24 (1.06) | 6.13 (0.653) | 20.1 (5.32) | 77.9 (15.5) | 109 (29.6) | 157 (56.8) | 148 (18.2) | 102 (36.1) | 131 (51.3) | 18.6 (3.94) | 67.1 (14.9) | 61.7 (13.4) | 71.5 (51.7) | 62.5 (20.2) | 48.9 (19.8) | 120 (6.24) | 131 (52.7) | 89.3 (2.71)
  Cycle 1 Day 1: 1 hour: number analyzed (Participants) | 3 | 4 | 7 | 8 | 12 | 3 | 5 | 43 | 27 | 2 | 6 | 33 | 23 | 24 | 36 | 3 | 20 | 1
  Cycle 1 Day 1: 1 hour | 1.61 (0.265) | 5.67 (1.61) | 16.6 (3.84) | 58.8 (25.3) | 112 (24.5) | 132 (33.0) | 135 (33.9) | 101 (32.3) | 117 (19.9) | 17.4 (5.33) | 50.0 (22.3) | 56.3 (11.2) | 61.6 (25.5) | 57.5 (17.9) | 49.9 (37.0) | 120 (22.0) | 121 (32.2) | 86.3 (NA) — Standard Deviation could not be calculated for 1 participant.
  Cycle 1 Day 1: 2 hours: number analyzed (Participants) | 3 | 4 | 7 | 8 | 12 | 3 | 5 | 45 | 27 | 3 | 6 | 34 | 24 | 24 | 35 | 3 | 20 | 2
  Cycle 1 Day 1: 2 hours | 0.965 (0.0894) | 3.83 (1.01) | 12.3 (2.80) | 44.0 (18.5) | 83.0 (19.6) | 98.9 (21.8) | 100 (27.1) | 77.4 (21.5) | 97.6 (21.7) | 14.0 (2.74) | 38.7 (17.4) | 42.5 (9.20) | 43.6 (11.5) | 42.6 (13.8) | 34.0 (18.8) | 94.9 (19.7) | 93.5 (30.7) | 70.7 (5.51)
  Cycle 1 Day 1: 4 hours: number analyzed (Participants) | 5 | 3 | 7 | 8 | 12 | 3 | 6 | 45 | 27 | 3 | 6 | 35 | 24 | 26 | 37 | 3 | 20 | 2
  Cycle 1 Day 1: 4 hours | 0.142 (0.318) | 1.87 (0.710) | 6.97 (2.25) | 25.2 (11.7) | 51.4 (15.9) | 57.4 (11.9) | 62.1 (26.5) | 50.1 (16.2) | 66.4 (15.9) | 8.74 (1.50) | 21.9 (7.94) | 25.6 (5.22) | 27.6 (7.91) | 26.4 (8.67) | 22.5 (13.6) | 63.8 (12.3) | 59.7 (15.5) | 48.9 (12.6)
  Cycle 1 Day 1: 8 hours: number analyzed (Participants) | 5 | 4 | 6 | 8 | 11 | 3 | 6 | 43 | 26 | 2 | 6 | 32 | 25 | 25 | 32 | 3 | 20 | 1
  Cycle 1 Day 1: 8 hours | 0.00 (0.00) | 0.453 (0.314) | 2.55 (1.27) | 10.0 (4.85) | 21.6 (7.61) | 24.9 (9.77) | 31.2 (16.9) | 31.8 (28.9) | 32.5 (7.83) | 4.49 (1.26) | 9.63 (4.37) | 10.2 (2.88) | 10.8 (4.41) | 10.8 (4.29) | 11.8 (11.9) | 27.7 (6.94) | 30.2 (8.92) | 18.7 (NA) — Standard Deviation could not be calculated for 1 participant.
  Cycle 1 Day 1: 16 hours: number analyzed (Participants) | 5 | 4 | 5 | 4 | 4 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Cycle 1 Day 1: 16 hours | 0.00 (0.00) | 0.00 (0.00) | 0.522 (0.641) | 1.50 (1.20) | 7.27 (4.49) |  |  |  |  |  | 0.00 (NA) — Standard Deviation could not be calculated for 1 participant. |  |  | 4.95 (NA) — Standard Deviation could not be calculated for 1 participant. |  |  |  |
  Cycle 1 Day 1: 24 hours: number analyzed (Participants) | 5 | 4 | 7 | 8 | 11 | 2 | 6 | 44 | 26 | 2 | 5 | 31 | 24 | 25 | 37 | 3 | 20 | 2
  Cycle 1 Day 1: 24 hours | 0.00 (0.00) | 0.00 (0.00) | 0.106 (0.280) | 1.19 (0.633) | 2.95 (1.61) | 3.21 (0.253) | 5.18 (4.20) | 3.64 (1.90) | 3.53 (1.25) | 0.498 (0.704) | 1.46 (0.803) | 1.64 (1.44) | 1.64 (1.42) | 1.29 (0.749) | 2.94 (6.88) | 4.49 (2.06) | 13.8 (43.0) | 3.45 (1.59)
  Cycle 1 Day 5: 0 hour: number analyzed (Participants) | 5 | 4 | 7 | 7 | 10 | 3 | 4 | 37 | 20 | 3 | 6 | 33 | 20 | 22 | 37 | 3 | 17 | 2
  Cycle 1 Day 5: 0 hour | 0.00 (0.00) | 0.00 (0.00) | 0.104 (0.276) | 0.619 (0.462) | 2.36 (2.29) | 1.59 (0.692) | 1.67 (0.531) | 1.51 (0.654) | 1.96 (0.987) | 0.209 (0.361) | 0.416 (0.538) | 1.10 (0.965) | 2.16 (3.95) | 0.933 (0.529) | 3.90 (9.89) | 2.03 (0.979) | 2.67 (2.06) | 1.92 (0.336)
  Cycle 1 Day 5: 0.5 hour: number analyzed (Participants) | 4 | 3 | 6 | 5 | 8 | 3 | 4 | 32 | 16 | 3 | 5 | 30 | 17 | 20 | 31 | 2 | 16 | 2
  Cycle 1 Day 5: 0.5 hour | 2.00 (0.238) | 6.00 (1.45) | 20.1 (8.08) | 71.3 (14.0) | 111 (26.0) | 112 (14.6) | 104 (13.0) | 85.1 (28.1) | 101 (29.2) | 19.5 (3.90) | 49.5 (19.7) | 58.3 (25.3) | 63.6 (41.8) | 61.1 (30.1) | 51.8 (29.6) | 118 (2.15) | 111 (42.4) | 104 (1.86)
  Cycle 1 Day 5: 1 hour: number analyzed (Participants) | 3 | 3 | 7 | 6 | 8 | 3 | 3 | 35 | 15 | 2 | 5 | 31 | 19 | 21 | 31 | 2 | 16 | 1
  Cycle 1 Day 5: 1 hour | 1.55 (0.245) | 5.28 (1.07) | 13.8 (7.79) | 48.9 (26.6) | 87.6 (14.7) | 98.4 (10.5) | 70.3 (9.27) | 78.0 (29.5) | 83.8 (14.8) | 18.9 (2.50) | 45.6 (22.3) | 47.2 (12.7) | 47.3 (12.2) | 41.9 (11.7) | 45.0 (28.2) | 105 (14.3) | 102 (29.5) | 89.8 (NA) — Standard Deviation could not be calculated for 1 participant.
  Cycle 1 Day 5: 2 hours: number analyzed (Participants) | 3 | 3 | 7 | 7 | 9 | 3 | 4 | 33 | 14 | 2 | 5 | 31 | 19 | 22 | 32 | 2 | 16 | 2
  Cycle 1 Day 5: 2 hours | 0.909 (0.164) | 3.53 (1.10) | 9.26 (5.76) | 30.1 (18.1) | 65.2 (22.1) | 66.4 (6.97) | 66.2 (15.1) | 57.8 (20.2) | 61.0 (14.3) | 13.1 (0.626) | 31.8 (17.0) | 30.6 (9.57) | 31.8 (9.39) | 27.4 (9.80) | 39.6 (38.3) | 65.1 (0.651) | 71.1 (23.8) | 66.5 (4.01)
  Cycle 1 Day 5: 4 hours: number analyzed (Participants) | 5 | 3 | 7 | 7 | 9 | 2 | 4 | 36 | 14 | 3 | 5 | 33 | 19 | 22 | 32 | 2 | 16 | 2
  Cycle 1 Day 5: 4 hours | 0.00 (0.00) | 1.17 (0.450) | 4.17 (3.72) | 12.9 (7.19) | 32.0 (14.0) | 29.1 (7.92) | 28.0 (14.0) | 39.4 (43.2) | 30.3 (6.20) | 6.18 (0.687) | 13.1 (11.7) | 13.2 (5.51) | 17.2 (18.5) | 13.0 (7.01) | 17.7 (16.2) | 28.4 (1.42) | 32.4 (13.5) | 33.4 (7.99)
  Cycle 1 Day 5: 8 hours: number analyzed (Participants) | 5 | 4 | 7 | 7 | 8 | 2 | 4 | 28 | 14 | 3 | 5 | 32 | 17 | 19 | 26 | 2 | 17 | 2
  Cycle 1 Day 5: 8 hours | 0.00 (0.00) | 0.00 (0.00) | 1.16 (1.31) | 3.25 (1.84) | 6.67 (2.74) | 6.68 (1.85) | 5.06 (1.68) | 6.78 (3.25) | 6.33 (2.04) | 1.86 (0.257) | 3.39 (3.39) | 3.41 (1.66) | 4.85 (3.63) | 3.26 (1.32) | 7.80 (12.3) | 20.2 (18.7) | 8.60 (5.71) | 7.22 (0.698)
  Cycle 1 Day 5: 16 hours: number analyzed (Participants) | 5 | 4 | 4 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 1 Day 5: 16 hours | 0.00 (0.00) | 0.158 (0.316) | 0.244 (0.488) | 0.625 (0.586) | 1.65 (0.707) |  |  |  |  |  |  |  |  |  |  |  |  |
  Cycle 1 Day 5: 24 hours: number analyzed (Participants) | 5 | 4 | 4 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 1 Day 5: 24 hours | 0.00 (0.00) | 0.00 (0.00) | 0.147 (0.294) | 0.221 (0.382) | 1.38 (0.631) |  |  |  |  |  |  |  |  |  |  |  |  |
  Cycle 1 Day 5: 72 hours: number analyzed (Participants) | 5 | 4 | 4 | 6 | 8 | 2 | 3 | 8 | 7 | 0 | 0 | 0 | 4 | 7 | 5 | 0 | 2 | 1
  Cycle 1 Day 5: 72 hours | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.498 (0.596) | 0.824 (0.333) | 0.664 (0.597) | 0.623 (0.973) | 0.538 (0.383) |  |  |  | 0.210 (0.419) | 0.103 (0.273) | 0.00 (0.00) |  | 0.610 (0.00778) | 0.989 (NA) — Standard Deviation could not be calculated for 1 participant.
  Cycle 2 Day 1: 0 hour: number analyzed (Participants) | 4 | 4 | 6 | 7 | 9 | 3 | 4 | 42 | 23 | 3 | 5 | 31 | 23 | 20 | 38 | 3 | 17 | 2
  Cycle 2 Day 1: 0 hour | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 8.24 (24.7) | 0.00 (0.00) | 0.00 (0.00) | 2.11 (13.7) | 0.120 (0.410) | 0.00 (0.00) | 0.00 (0.00) | 0.0170 (0.0945) | 0.00 (0.00) | 2.10 (9.24) | 0.00 (0.00) | 0.00 (0.00) | 0.372 (1.36) | 0.00 (0.00)
  Cycle 2 Day 1: 0.5 hour: number analyzed (Participants) | 4 | 1 | 6 | 5 | 4 | 3 | 3 | 36 | 22 | 2 | 5 | 26 | 22 | 19 | 34 | 3 | 16 | 0
  Cycle 2 Day 1: 0.5 hour | 1.80 (0.590) | 5.42 (NA) — Standard Deviation could not be calculated for 1 participant. | 20.7 (6.83) | 72.2 (13.0) | 105 (23.9) | 113 (15.1) | 121 (40.4) | 174 (372) | 123 (31.7) | 15.8 (2.82) | 56.3 (9.99) | 57.8 (15.4) | 79.6 (93.1) | 55.7 (22.7) | 51.1 (28.0) | 113 (16.8) | 137 (47.3) |
  Cycle 2 Day 1: 1 hour: number analyzed (Participants) | 2 | 4 | 6 | 5 | 6 | 3 | 3 | 39 | 21 | 1 | 6 | 29 | 22 | 20 | 34 | 3 | 17 | 2
  Cycle 2 Day 1: 1 hour | 1.36 (0.646) | 4.84 (0.806) | 17.3 (5.46) | 58.3 (11.8) | 94.6 (14.3) | 105 (27.7) | 102 (33.2) | 93.3 (34.9) | 106 (30.3) | 13.7 (NA) — Standard Deviation could not be calculated for 1 participant. | 48.2 (13.7) | 51.5 (10.0) | 54.2 (14.2) | 47.8 (13.0) | 43.0 (27.4) | 117 (17.2) | 114 (29.2) | 120 (5.86)
  Cycle 2 Day 1: 2 hours: number analyzed (Participants) | 3 | 4 | 6 | 6 | 7 | 3 | 3 | 40 | 22 | 2 | 6 | 30 | 23 | 20 | 34 | 3 | 17 | 2
  Cycle 2 Day 1: 2 hours | 0.889 (0.174) | 3.43 (0.797) | 12.6 (4.40) | 44.9 (14.5) | 74.5 (18.2) | 76.9 (23.3) | 85.9 (26.8) | 76.7 (26.5) | 87.9 (23.5) | 11.3 (1.39) | 35.6 (8.32) | 38.8 (9.33) | 38.3 (11.1) | 37.1 (10.5) | 35.6 (30.6) | 92.6 (16.1) | 84.4 (24.6) | 89.7 (5.33)
  Cycle 2 Day 1: 4 hours: number analyzed (Participants) | 4 | 4 | 6 | 6 | 7 | 3 | 3 | 39 | 22 | 3 | 6 | 30 | 23 | 20 | 35 | 3 | 17 | 2
  Cycle 2 Day 1: 4 hours | 0.00 (0.00) | 1.31 (0.422) | 7.16 (3.53) | 27.8 (10.6) | 45.1 (14.0) | 50.5 (16.2) | 52.5 (15.8) | 46.8 (16.5) | 57.1 (14.9) | 7.00 (0.412) | 19.5 (4.90) | 25.1 (12.7) | 24.0 (7.15) | 21.4 (8.75) | 24.1 (19.1) | 54.9 (6.38) | 54.7 (16.7) | 58.0 (8.50)
  Cycle 2 Day 1: 8 hours: number analyzed (Participants) | 4 | 4 | 5 | 6 | 7 | 3 | 3 | 40 | 21 | 1 | 5 | 30 | 20 | 16 | 32 | 3 | 17 | 2
  Cycle 2 Day 1: 8 hours | 0.00 (0.00) | 0.00 (0.00) | 2.32 (1.45) | 9.29 (4.62) | 16.5 (7.44) | 18.7 (9.48) | 24.9 (13.1) | 26.8 (35.4) | 24.1 (8.09) | 2.51 (NA) — Standard Deviation could not be calculated for 1 participant. | 8.66 (4.83) | 7.91 (3.47) | 8.85 (3.92) | 7.40 (3.67) | 12.8 (18.3) | 24.3 (3.79) | 24.0 (11.5) | 26.4 (6.55)
  Cycle 2 Day 1: 16 hours: number analyzed (Participants) | 4 | 4 | 3 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  Cycle 2 Day 1: 16 hours | 0.00 (0.00) | 0.00 (0.00) | 0.405 (0.701) | 2.47 (2.14) | 4.24 (3.60) |  |  |  |  |  |  |  |  | 1.97 (NA) — Standard Deviation could not be calculated for 1 participant. | 1.69 (NA) — Standard Deviation could not be calculated for 1 participant. |  |  |
  Cycle 2 Day 1: 24 hours: number analyzed (Participants) | 4 | 4 | 6 | 6 | 7 | 3 | 3 | 40 | 22 | 2 | 6 | 28 | 20 | 19 | 35 | 3 | 15 | 2
  Cycle 2 Day 1: 24 hours | 0.00 (0.00) | 0.205 (0.410) | 0.219 (0.342) | 0.940 (0.561) | 2.11 (1.45) | 1.81 (1.30) | 2.51 (1.19) | 2.03 (1.69) | 1.95 (0.854) | 0.00 (0.00) | 0.737 (0.518) | 1.06 (1.06) | 1.16 (0.777) | 1.15 (1.40) | 4.96 (11.7) | 3.16 (1.58) | 2.98 (1.51) | 3.19 (1.10)
  Cycle 2 Day 5: 0 hour: number analyzed (Participants) | 3 | 4 | 6 | 5 | 10 | 2 | 3 | 40 | 21 | 3 | 6 | 27 | 22 | 18 | 37 | 2 | 16 | 2
  Cycle 2 Day 5: 0 hour | 0.00 (0.00) | 0.00 (0.00) | 0.0868 (0.213) | 0.914 (0.614) | 1.36 (0.589) | 2.24 (1.46) | 2.36 (1.11) | 1.58 (0.653) | 1.72 (0.599) | 0.180 (0.312) | 0.756 (0.786) | 2.14 (6.54) | 0.922 (0.670) | 1.01 (1.71) | 4.17 (8.72) | 1.45 (0.417) | 2.17 (1.46) | 1.86 (0.354)
  Cycle 2 Day 5: 0.5 hour: number analyzed (Participants) | 2 | 3 | 4 | 2 | 6 | 2 | 3 | 34 | 19 | 2 | 5 | 23 | 20 | 19 | 33 | 2 | 15 | 1
  Cycle 2 Day 5: 0.5 hour | 1.92 (0.296) | 6.06 (0.454) | 17.2 (3.44) | 69.1 (16.8) | 93.9 (22.2) | 98.8 (34.7) | 91.2 (40.2) | 153 (300) | 101 (18.6) | 13.4 (3.07) | 44.3 (9.53) | 64.2 (60.1) | 58.8 (38.5) | 52.7 (14.4) | 56.7 (31.1) | 100 (20.0) | 100 (28.8) | 103 (NA) — Standard Deviation could not be calculated for 1 participant.
  Cycle 2 Day 5: 1 hour: number analyzed (Participants) | 2 | 4 | 6 | 3 | 7 | 2 | 3 | 33 | 19 | 2 | 6 | 22 | 20 | 19 | 31 | 2 | 14 | 2
  Cycle 2 Day 5: 1 hour | 1.44 (0.260) | 4.82 (0.794) | 14.7 (3.80) | 44.9 (18.3) | 84.8 (23.7) | 90.5 (16.3) | 78.4 (39.9) | 94.8 (104) | 83.4 (19.4) | 16.8 (5.53) | 33.8 (7.91) | 69.8 (124) | 42.7 (12.9) | 42.3 (15.5) | 48.1 (28.2) | 86.3 (15.0) | 90.9 (24.6) | 89.7 (4.66)
  Cycle 2 Day 5: 2 hours: number analyzed (Participants) | 2 | 4 | 6 | 4 | 7 | 2 | 3 | 34 | 19 | 2 | 6 | 22 | 20 | 19 | 29 | 2 | 14 | 2
  Cycle 2 Day 5: 2 hours | 0.988 (0.0219) | 2.84 (0.751) | 9.09 (3.13) | 29.9 (12.3) | 58.4 (19.3) | 59.0 (6.87) | 49.9 (15.2) | 55.3 (20.9) | 62.0 (17.8) | 10.3 (4.44) | 21.3 (4.81) | 28.6 (9.10) | 29.9 (9.94) | 28.5 (9.68) | 36.7 (27.9) | 57.6 (10.5) | 59.9 (19.7) | 67.3 (4.50)
  Cycle 2 Day 5: 4 hours: number analyzed (Participants) | 3 | 4 | 6 | 4 | 7 | 2 | 3 | 35 | 19 | 3 | 6 | 25 | 21 | 19 | 34 | 2 | 15 | 2
  Cycle 2 Day 5: 4 hours | 0.00 (0.00) | 1.13 (0.471) | 4.18 (1.98) | 14.9 (6.75) | 27.1 (10.4) | 24.2 (2.26) | 24.3 (11.6) | 27.6 (8.71) | 29.1 (10.4) | 6.40 (2.13) | 8.11 (2.77) | 12.0 (4.47) | 14.8 (6.00) | 13.3 (5.22) | 25.2 (32.6) | 29.8 (2.81) | 30.8 (12.5) | 34.7 (8.12)
  Cycle 2 Day 5: 8 hours: number analyzed (Participants) | 3 | 4 | 6 | 5 | 7 | 2 | 2 | 29 | 18 | 3 | 6 | 25 | 17 | 16 | 27 | 2 | 15 | 2
  Cycle 2 Day 5: 8 hours | 0.00 (0.00) | 0.00 (0.00) | 1.27 (0.509) | 3.89 (1.58) | 6.93 (3.91) | 5.74 (0.0933) | 7.51 (3.23) | 7.94 (6.53) | 6.49 (2.96) | 1.47 (0.445) | 28.2 (64.5) | 3.33 (1.87) | 3.99 (1.69) | 3.94 (1.97) | 12.2 (19.7) | 4.98 (1.92) | 9.78 (5.22) | 8.47 (3.87)
  Cycle 2 Day 5: 16 hours: number analyzed (Participants) | 3 | 4 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 2 Day 5: 16 hours | 0.00 (0.00) | 0.00 (0.00) | 0.218 (0.378) | 1.15 (0.687) | 1.64 (0.597) |  |  |  |  |  |  |  |  |  |  |  |  |
  Cycle 2 Day 5: 24 hours: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 2 Day 5: 24 hours | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.631 (0.630) | 1.38 (0.697) |  |  |  |  |  |  |  |  |  |  |  |  |
  Cycle 2 Day 5: 72 hours: number analyzed (Participants) | 3 | 3 | 2 | 3 | 7 | 3 | 2 | 6 | 11 | 0 | 0 | 0 | 1 | 6 | 4 | 0 | 2 | 1
  Cycle 2 Day 5: 72 hours | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.200 (0.347) | 0.488 (0.376) | 0.611 (0.625) | 1.57 (0.584) | 0.578 (0.475) | 0.396 (0.450) |  |  |  | 0.00 (NA) — Standard Deviation could not be calculated for 1 participant. | 0.00 (0.00) | 0.00 (0.00) |  | 1.17 (0.409) | 0.741 (NA) — Standard Deviation could not be calculated for 1 participant.
  Cycle 2 Day 5: 240 hours: number analyzed (Participants) | 3 | 2 | 3 | 5 | 6 | 2 | 3 | 10 | 12 | 0 | 0 | 2 | 2 | 10 | 6 | 1 | 7 | 0
  Cycle 2 Day 5: 240 hours | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) |  |  | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (NA) — Standard Deviation could not be calculated for 1 participant. | 0.00 (0.00) |

6. Secondary Outcome: Parts A, B and C: Area Under Concentration From Time Zero to the Last Quantifiable Concentration (AUClast) of Nemvaleukin Alfa
Description: Cycle 1 length = 14 days for Part A and 21 days for Part B and C; Cycle 2 length= 21 days for all parts.
Time Frame: as for outcome 5
Population: The PK population consisted of all participants who received at least 1 dose of nemvaleukin alfa and had at least 1 measurable serum concentration of nemvaleukin alfa at any scheduled PK time point. Here, "overall number of participants analyzed" signifies participants who were evaluable for this outcome measure and "number analyzed" signifies participants who were evaluable at specified timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Groups:
- Part C, Combination Therapy, Cohort 1: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg: Participants with PD-1/L1 unapproved tumor types (PD-1/L1 treatment naive) received nemvaleukin alfa 3 mcg/kg IV infusion administration daily from Days 1 to 5 in combination with pembrolizumab 200 mg IV infusion on Day 1 in each Cycle (cycle length = 21 days) for a maximum of 2 years for as long as the participant appeared to be deriving clinical benefit (i.e., objective response or SD) and had tolerated therapy well. Participants could continue nemvaleukin alfa as monotherapy beyond the maximum of 2 years of treatment by switching to monotherapy at the joint discretion of the Investigator and Sponsor and if they did not meet any other criteria for discontinuation.
Arm/Group | Part A, Dose Escalation: Nemvaleukin Alfa 0.1 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 0.3 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 1 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 3 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 6 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 8 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 10 mcg/kg | Part B, Dose Expansion, Melanoma: Nemvaleukin Alfa 6 mcg/kg | Part B, Dose Expansion, RCC: Nemvaleukin Alfa 6 mcg/kg | Part C, Combination Therapy, Safety Run-in: Nemvaleukin Alfa 1 mcg/kg | Part C, Combination Therapy, Safety Run-in: Nemvaleukin Alfa 3 mcg/kg | Part C, Combination Therapy, Cohort 1: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 2: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 3: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Rollover, Cohort 4: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 5: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 6: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 7: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg
Number analyzed (Participants) | 5 | 4 | 6 | 8 | 12 | 3 | 6 | 44 | 27 | 3 | 6 | 34 | 24 | 26 | 36 | 3 | 20 | 2
hour*nanogram per milliliter (h*ng/mL)
  Cycle 1 Day 1 | 2.96 (53.1) | 17.0 (35.6) | 66.5 (36.5) | 195 (252.1) | 557 (28.7) | 616 (42.3) | 719 (39.7) | 608 (30.1) | 723 (23.2) | 84.1 (39.5) | 248 (23.4) | 286 (22.1) | 296 (35.0) | 276 (31.4) | 222 (77.2) | 698 (21.7) | 715 (37.6) | 543 (25.0)
  Cycle 1 Day 5: number analyzed (Participants) | 5 | 4 | 6 | 7 | 9 | 3 | 4 | 35 | 15 | 3 | 5 | 33 | 19 | 22 | 33 | 2 | 16 | 2
  Cycle 1 Day 5 | 2.52 (17.3) | 14.4 (23.6) | 48.2 (55.9) | 106 (205.5) | 379 (46.0) | 323 (84.1) | 346 (47.8) | 292 (61.4) | 312 (40.6) | 56.7 (18.8) | 121 (68.5) | 143 (26.2) | 158 (41.6) | 130 (40.5) | 139 (53.4) | 343 (6.8) | 368 (56.7) | 393 (45.8)
  Cycle 2 Day 1: number analyzed (Participants) | 4 | 3 | 6 | 6 | 7 | 3 | 3 | 41 | 22 | 2 | 6 | 29 | 23 | 20 | 35 | 3 | 17 | 1
  Cycle 2 Day 1 | 2.47 (32.4) | 15.3 (45.4) | 69.2 (50.3) | 274 (39.0) | 478 (30.7) | 512 (35.6) | 573 (36.8) | 517 (44.5) | 594 (25.9) | 56.1 (12.9) | 195 (50.1) | 235 (30.8) | 243 (41.5) | 212 (39.6) | 224 (85.0) | 625 (12.5) | 562 (33.5) | 590 (NA) — Geometric Coefficient of Variation could not be calculated for 1 participant.
  Cycle 2 Day 5: number analyzed (Participants) | 3 | 4 | 5 | 5 | 7 | 2 | 3 | 35 | 19 | 3 | 6 | 25 | 21 | 17 | 32 | 2 | 15 | 2
  Cycle 2 Day 5 | 2.61 (16.6) | 11.5 (18.4) | 40.8 (21.2) | 167 (51.5) | 361 (50.4) | 439 (3.5) | 312 (131.0) | 287 (60.9) | 329 (45.3) | 52.0 (18.5) | 120 (72.3) | 135 (54.3) | 134 (35.4) | 128 (36.6) | 153 (73.4) | 275 (15.0) | 346 (43.9) | 413 (57.6)

7. Secondary Outcome: Parts A, B and C: Maximum Observed Serum Concentration (Cmax) of Nemvaleukin Alfa
Description: Cycle 1 length = 14 days for Part A and 21 days for Part B and C; Cycle 2 length= 21 days for all parts.
Time Frame: as for outcome 5
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliters (ng/mL)
Arm/Group | Part A, Dose Escalation: Nemvaleukin Alfa 0.1 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 0.3 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 1 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 3 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 6 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 8 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 10 mcg/kg | Part B, Dose Expansion, Melanoma: Nemvaleukin Alfa 6 mcg/kg | Part B, Dose Expansion, RCC: Nemvaleukin Alfa 6 mcg/kg | Part C, Combination Therapy, Safety Run-in: Nemvaleukin Alfa 1 mcg/kg | Part C, Combination Therapy, Safety Run-in: Nemvaleukin Alfa 3 mcg/kg | Part C, Combination Therapy, Cohort 1: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 2: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 3: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Rollover, Cohort 4: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 5: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 6: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 7: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg
Number analyzed (Participants) | 5 | 4 | 6 | 8 | 11 | 3 | 6 | 44 | 27 | 3 | 6 | 34 | 23 | 25 | 36 | 3 | 18 | 2
nanograms per milliliters (ng/mL)
  Cycle 1 Day 1 | 2.09 (41.4) | 6.72 (21.3) | 20.5 (26.8) | 47.6 (177.8) | 113 (33.7) | 151 (36.7) | 157 (19.4) | 99.4 (40.8) | 124 (34.2) | 18.1 (15.4) | 65.6 (24.4) | 61.4 (22.8) | 57.5 (86.5) | 59.5 (32.6) | 45.8 (48.8) | 131 (15.8) | 133 (31.7) | 89.3 (3.0)
  Cycle 1 Day 5: number analyzed (Participants) | 5 | 4 | 6 | 8 | 9 | 3 | 4 | 36 | 15 | 3 | 5 | 33 | 19 | 22 | 33 | 2 | 16 | 2
  Cycle 1 Day 5 | 1.99 (10.3) | 6.36 (24.5) | 37.4 (19.2) | 41.8 (178.7) | 108 (22.5) | 112 (13.5) | 104 (12.5) | 82.1 (32.3) | 95.1 (33.8) | 19.2 (21.7) | 46.5 (41.6) | 55.8 (37.5) | 53.1 (57.9) | 54.4 (51.8) | 47.0 (40.1) | 118 (1.8) | 101 (51.5) | 104 (1.8)
  Cycle 2 Day 1: number analyzed (Participants) | 4 | 2 | 6 | 8 | 6 | 3 | 3 | 40 | 22 | 2 | 6 | 27 | 23 | 20 | 35 | 3 | 17 | 1
  Cycle 2 Day 1 | 1.72 (35.1) | 5.34 (2.2) | 19.8 (32.3) | 65.3 (27.5) | 113 (24.7) | 112 (13.0) | 116 (33.1) | 108 (86.7) | 119 (27.6) | 15.6 (18.1) | 52.9 (21.9) | 55.8 (26.9) | 58.1 (81.2) | 55.6 (31.4) | 47.2 (47.7) | 112 (15.3) | 128 (30.6) | 124 (NA) — Geometric Coefficient of Variation could not be calculated for 1 participant.
  Cycle 2 Day 5: number analyzed (Participants) | 3 | 4 | 6 | 5 | 7 | 2 | 3 | 35 | 19 | 3 | 6 | 24 | 21 | 19 | 32 | 2 | 15 | 2
  Cycle 2 Day 5 | 1.90 (11.0) | 6.39 (12.7) | 16.7 (18.5) | 52.9 (48.1) | 97.4 (29.0) | 95.7 (37.0) | 83.8 (57.4) | 103 (69.5) | 99.6 (18.3) | 14.6 (24.0) | 40.8 (26.9) | 50.3 (67.9) | 51.7 (52.0) | 51.0 (25.9) | 49.8 (52.6) | 99.2 (20.3) | 96.6 (29.7) | 94.4 (12.5)

8. Secondary Outcome: Parts A, B and C: Time to Reach Cmax (Tmax) of Nemvaleukin Alfa
Description: Cycle 1 length = 14 days for Part A and 21 days for Part B and C; Cycle 2 length= 21 days for all parts.
Time Frame: as for outcome 5
Population: as for outcome 6
Measure: Median (Full Range); unit: hours
Arm/Group | Part A, Dose Escalation: Nemvaleukin Alfa 0.1 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 0.3 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 1 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 3 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 6 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 8 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 10 mcg/kg | Part B, Dose Expansion, Melanoma: Nemvaleukin Alfa 6 mcg/kg | Part B, Dose Expansion, RCC: Nemvaleukin Alfa 6 mcg/kg | Part C, Combination Therapy, Safety Run-in: Nemvaleukin Alfa 1 mcg/kg | Part C, Combination Therapy, Safety Run-in: Nemvaleukin Alfa 3 mcg/kg | Part C, Combination Therapy, Cohort 1: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 2: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 3: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Rollover, Cohort 4: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 5: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 6: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 7: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg
Number analyzed (Participants) | 5 | 4 | 6 | 8 | 11 | 3 | 6 | 44 | 27 | 3 | 6 | 34 | 23 | 25 | 36 | 3 | 18 | 2
hours
  Cycle 1 Day 1 | 0.60 [0.57 to 0.83] | 0.63 [0.52 to 0.73] | 0.55 [0.50 to 0.78] | 0.57 [0.50 to 0.75] | 0.57 [0.50 to 0.70] | 0.57 [0.53 to 0.57] | 0.51 [0.50 to 0.62] | 0.52 [0.50 to 0.75] | 0.50 [0.50 to 0.67] | 0.75 [0.57 to 0.98] | 0.73 [0.58 to 0.75] | 0.55 [0.48 to 1.00] | 0.55 [0.50 to 0.73] | 0.52 [0.40 to 0.63] | 0.50 [0.50 to 0.82] | 0.50 [0.50 to 0.67] | 0.53 [0.45 to 1.00] | 0.78 [0.50 to 1.07]
  Cycle 1 Day 5: number analyzed (Participants) | 5 | 4 | 6 | 7 | 9 | 3 | 4 | 36 | 15 | 3 | 5 | 33 | 19 | 22 | 33 | 2 | 16 | 2
  Cycle 1 Day 5 | 0.70 [0.50 to 0.80] | 0.60 [0.48 to 0.82] | 0.54 [0.50 to 0.80] | 0.55 [0.50 to 0.67] | 0.58 [0.53 to 0.73] | 0.53 [0.53 to 0.58] | 0.53 [0.50 to 0.68] | 0.51 [0.50 to 0.80] | 0.50 [0.43 to 0.58] | 0.58 [0.55 to 0.72] | 0.73 [0.55 to 0.77] | 0.57 [0.50 to 1.00] | 0.53 [0.30 to 0.85] | 0.55 [0.48 to 0.68] | 0.50 [0.50 to 0.75] | 0.58 [0.58 to 0.58] | 0.52 [0.45 to 0.63] | 0.83 [0.57 to 1.08]
  Cycle 2 Day 1: number analyzed (Participants) | 4 | 2 | 6 | 6 | 6 | 3 | 3 | 44 | 22 | 2 | 6 | 27 | 23 | 20 | 35 | 3 | 17 | 1
  Cycle 2 Day 1 | 0.67 [0.58 to 0.80] | 0.73 [0.72 to 0.75] | 0.53 [0.50 to 0.58] | 0.55 [0.50 to 0.87] | 0.58 [0.55 to 0.73] | 0.53 [0.52 to 0.58] | 0.52 [0.50 to 0.63] | 0.50 [0.50 to 0.77] | 0.50 [0.50 to 0.60] | 0.71 [0.60 to 0.82] | 0.68 [0.57 to 0.80] | 0.55 [0.50 to 1.00] | 0.53 [0.47 to 1.00] | 0.53 [0.50 to 0.58] | 0.50 [0.50 to 0.77] | 0.55 [0.50 to 0.58] | 0.52 [0.48 to 0.68] | 1.00 [1.00 to 1.00]
  Cycle 2 Day 5: number analyzed (Participants) | 3 | 4 | 5 | 5 | 7 | 2 | 3 | 35 | 19 | 3 | 6 | 24 | 21 | 19 | 32 | 2 | 15 | 2
  Cycle 2 Day 5 | 0.63 [0.55 to 0.80] | 0.57 [0.50 to 0.68] | 0.55 [0.50 to 0.75] | 0.68 [0.52 to 1.58] | 0.60 [0.50 to 0.75] | 0.58 [0.58 to 0.58] | 0.52 [0.50 to 0.52] | 0.50 [0.50 to 0.77] | 0.50 [0.50 to 0.67] | 0.72 [0.55 to 0.73] | 0.68 [0.58 to 0.78] | 0.55 [0.52 to 1.00] | 0.55 [0.50 to 1.08] | 0.50 [0.48 to 0.62] | 0.50 [0.50 to 0.62] | 0.56 [0.50 to 0.62] | 0.52 [0.50 to 0.58] | 0.77 [0.53 to 1.00]

9. Secondary Outcome: Parts A, B, and C: Proportion of Positive Anti-Nemvaleukin Alfa Antibodies (ADA)
Description: Overall proportion was calculated as: Number of participants (overall positive)/total number of participants in the cohort. Overall positive: Participants with at least 1 treatment-emergent ADA positive sample at any time during the treatment period.
Time Frame: From first dose of study drug up to 9 months (for Part A); up to 40.3 months (for Part B); up to 50.5 months (for Part C)
Population: Immunogenicity analysis set included all participants who received at least one dose of active study drug and had at least one post baseline blood sample collected to assess immunogenicity.
Measure: Number; unit: proportion of participants
Arm/Group | Part A, Dose Escalation: Nemvaleukin Alfa 0.1 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 0.3 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 1 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 3 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 6 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 8 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 10 mcg/kg | Part B, Dose Expansion, Melanoma: Nemvaleukin Alfa 6 mcg/kg | Part B, Dose Expansion, RCC: Nemvaleukin Alfa 6 mcg/kg | Part C, Combination Therapy, Safety Run-in: Nemvaleukin Alfa 1 mcg/kg | Part C, Combination Therapy, Safety Run-in: Nemvaleukin Alfa 3 mcg/kg | Part C, Combination Therapy, Cohort 1: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 2: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 3: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Rollover, Cohort 4: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 5: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 6: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 7: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg
Number analyzed (Participants) | 5 | 4 | 7 | 8 | 12 | 3 | 5 | 45 | 26 | 3 | 6 | 34 | 24 | 24 | 43 | 3 | 20 | 2
proportion of participants | 0.00 | 0.00 | 0.143 | 0.125 | 0.417 | 0.333 | 0.600 | 0.467 | 0.500 | 0.00 | 0.667 | 0.294 | 0.250 | 0.208 | 0.581 | 0.667 | 0.200 | 0.00

10. Secondary Outcome: Parts A, B, and C: Immune ORR (iORR) Based on Immune RECIST (iRECIST)
Description: iORR was defined as the percentage of participants with objective evidence of immune CR (iCR) or immune PR (iPR) based on iRECIST guidelines.
Time Frame: From first dose of study drug up to 9 months for Part A; up to 40.3 months for Part B; up to 50.5 months for Part C
Population: No data collection or analysis based on immune-related response criteria (irRC) and iRECIST was performed as iRECIST was implemented during the middle of the study conduct to replace irRC. However, no data was collected and analyzed for iRECIST either. Therefore, no data is available to report for this outcome measure.
Groups:
- Part C, Combination Therapy, Cohort 7: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg: Participants with SCCHN received nemvaleukin alfa 6 mcg/kg IV administration daily from Days 1 to 5 in combination with pembrolizumab 200 mg IV infusion on Day 1 in each Cycle (cycle length = 21 days) for a maximum of 2 years for as long as the participant appeared to be deriving clinical benefit (i.e., objective response or SD) and had tolerated therapy well. Participants could continue nemvaleukin alfa as monotherapy beyond the maximum of 2 years of treatment by switching to monotherapy at the joint discretion of the Investigator and Sponsor and if they did not meet any other criteria for discontinuation.
Arm/Group | Part A, Dose Escalation: Nemvaleukin Alfa 0.1 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 0.3 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 1 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 3 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 6 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 8 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 10 mcg/kg | Part B, Dose Expansion, Melanoma: Nemvaleukin Alfa 6 mcg/kg | Part B, Dose Expansion, RCC: Nemvaleukin Alfa 6 mcg/kg | Part C, Combination Therapy, Safety Run-in: Nemvaleukin Alfa 1 mcg/kg | Part C, Combination Therapy, Cohort 1 +Safety Run-in: Nemvaleukin Alfa 3 mcg/kg+Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 2: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 3: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Rollover, Cohort 4: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 5: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 6: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 7: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Parts A, B, and C: Disease Control Rate (DCR) Based on RECIST v.1.1
Description: Disease control rate was defined as the percentage of participants with objective evidence of CR, PR, or SD based on RECIST v.1.1. CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: From first dose of study drug up to 9 months for Part A; up to 40.3 months for Part B; up to 50.5 months for Part C
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Part A, Dose Escalation: Nemvaleukin 0.3 mcg/kg: Participants with advanced solid tumors received nemvaleukin alfa 0.3 mcg/kg IV infusion administration daily from Days 1 to 5 in Cycle 1 (Cycle length = 14 days) and then in Cycle 2 and subsequent cycles (each Cycle length = 21 days) until disease progression or the participant met any discontinuation criteria.
- Part C, Combination Therapy, Cohort 1+ Safety Run-in: Nemvaleukin Alfa 3 mcg/kg +Pembrolizumab 200mg: Participants with PD-1/L1 unapproved tumor types (PD-1/L1 treatment naive) received nemvaleukin alfa 3 mcg/kg IV infusion administration daily from Days 1 to 5 in combination with pembrolizumab 200 mg IV infusion on Day 1 in each Cycle (cycle length = 21 days) for a maximum of 2 years for as long as the participant appeared to be deriving clinical benefit (i.e., objective response or SD) and had tolerated therapy well. Participants could continue nemvaleukin alfa as monotherapy beyond the maximum of 2 years of treatment by switching to monotherapy at the joint discretion of the Investigator and Sponsor and if they did not meet any other criteria for discontinuation. The Safety Run-in for nemvaleukin alfa 3 mcg/kg was combined with Cohort 1 of Part C due to same dosing level and regimen.
Arm/Group | Part A, Dose Escalation: Nemvaleukin Alfa 0.1 mcg/kg | Part A, Dose Escalation: Nemvaleukin 0.3 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 1 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 3 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 6 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 8 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 10 mcg/kg | Part B, Dose Expansion, Melanoma: Nemvaleukin Alfa 6 mcg/kg | Part B, Dose Expansion, RCC: Nemvaleukin Alfa 6 mcg/kg | Part C, Combination Therapy, Safety Run-in: Nemvaleukin Alfa 1 mcg/kg | Part C, Combination Therapy, Cohort 1+ Safety Run-in: Nemvaleukin Alfa 3 mcg/kg +Pembrolizumab 200mg | Part C, Combination Therapy, Cohort 2: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 3: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Rollover, Cohort 4: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 5: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 6: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 7: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg
Number analyzed (Participants) | 4 | 4 | 5 | 5 | 9 | 3 | 4 | 46 | 22 | 3 | 36 | 22 | 21 | 39 | 3 | 18 | 2
percentage of participants | 0.0 [0.0 to 60.2] | 25.0 [0.6 to 80.6] | 20.0 [0.5 to 71.6] | 60.0 [14.7 to 94.7] | 33.3 [7.5 to 70.1] | 33.3 [0.8 to 90.6] | 25.0 [0.6 to 80.6] | 47.8 [32.9 to 63.1] | 50.0 [28.2 to 71.8] | 0.0 [0.0 to 70.8] | 30.6 [16.3 to 48.1] | 22.7 [7.8 to 45.4] | 47.6 [25.7 to 70.2] | 46.2 [30.1 to 62.8] | 66.7 [9.4 to 99.2] | 50.0 [26.0 to 74.0] | 100 [15.8 to 100.0]

12. Secondary Outcome: Parts A, B, and C: Immune DCR (iDCR) Based on iRECIST v1.1
Description: iDCR was defined as the percentage of participants with objective evidence of iCR, iPR (where iCR or iPR required confirmation), or immune stable disease (iSD) (where the iSD requires to occur at Cycle 4 or later).
Time Frame: From first dose of study drug up to 9 months for Part A; up to 40.3 months for Part B; up to 50.5 months for Part C
Population: No data collection or analysis based on irRC and iRECIST was performed as iRECIST was implemented during the middle of the study conduct to replace irRC. However, no data was collected and analyzed for iRECIST either. Therefore, no data is available to report for this outcome measure.
Groups:
- Part C, Combination Therapy, Cohort 2: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg: Participants with PD-1/L1 approved tumor types (PD-1/L1 treatment pretreated) received nemvaleukin alfa 3 mcg/kg infusion IV administration daily from Days 1 to 5 in combination with pembrolizumab 200 mg IV infusion on Day 1 in each Cycle (cycle length = 21 days) for a maximum of 2 years for as long as the participant appeared to be deriving clinical benefit (i.e., objective response or SD) and had tolerated therapy well. Participants could continue nemvaleukin alfa as monotherapy beyond the maximum of 2 years of treatment by switching to monotherapy at the joint discretion of the Investigator and Sponsor and if they did not meet any other criteria for discontinuation.
Arm/Group | Part A, Dose Escalation: Nemvaleukin Alfa 0.1 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 0.3 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 1 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 3 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 6 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 8 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 10 mcg/kg | Part B, Dose Expansion, Melanoma: Nemvaleukin Alfa 6 mcg/kg | Part B, Dose Expansion, RCC: Nemvaleukin Alfa 6 mcg/kg | Part C, Combination Therapy, Safety Run-in: Nemvaleukin Alfa 1 mcg/kg | Part C, Combination Therapy, Cohort 1 +Safety Run-in: Nemvaleukin Alfa 3 mcg/kg+Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 2: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 3: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Rollover, Cohort 4: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 5: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 6: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 7: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Parts B, and C: Duration of Response (DOR) Based on RECIST v1.1
Description: Duration of response was defined as the time from the first documentation of response (CR or PR) to the first documentation of objective tumor progression or death due to any cause. CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. PD: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: From the first documentation of response (CR or PR) to the first documentation of objective tumor progression or death due to any cause (up to 40.3 months for Part B and up to 50.5 months for Part C)
Population: The antitumor evaluable population consisted of participants who complete 2 cycles of therapy and had at least one follow-up scan. Here, "overall number of participants analyzed" signified participants who had CR or PR.
Measure: Median (95% Confidence Interval); unit: weeks
Groups:
- Part C, Combination Therapy, Rollover, Cohort 4: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg: Participants rollover from Parts A or B received nemvaleukin alfa 3 mcg/kg IV infusion administration daily from Days 1 to 5 in combination with pembrolizumab alfa 200 mg IV infusion on Day 1 in each Cycle (cycle length = 21 days) for a maximum of 2 years for as long as the participant appeared to be deriving clinical benefit (i.e., objective response or SD) and had tolerated therapy well. Participants could continue nemvaleukin alfa as monotherapy beyond the maximum of 2 years of treatment by switching to monotherapy at the joint discretion of the Investigator and Sponsor and if they did not meet any other criteria for discontinuation.
Arm/Group | Part B, Dose Expansion, Melanoma: Nemvaleukin Alfa 6 mcg/kg | Part B, Dose Expansion, RCC: Nemvaleukin Alfa 6 mcg/kg | Part C, Combination Therapy, Safety Run-in: Nemvaleukin Alfa 1 mcg/kg | Part C, Combination Therapy, Cohort 1 +Safety Run-in: Nemvaleukin Alfa 3 mcg/kg +Pembrolizumab 200mg | Part C, Combination Therapy, Cohort 2: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 3: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Rollover, Cohort 4: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 5: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 6: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 7: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg
Number analyzed (Participants) | 6 | 4 | 0 | 6 | 1 | 7 | 5 | 2 | 2 | 1
weeks | 18.43 [6.14 to NA] — Here, NA means upper limit of confidence interval could not be estimated due to insufficient events. | 28.86 [12.43 to NA] — Here, NA means upper limit of confidence interval could not be estimated due to insufficient events. |  | 35.14 [8.29 to 160.14] | NA [NA to NA] — Here, NA means median and confidence interval could not be estimated due to insufficient events. | 63.14 [6.86 to NA] — Here, NA means upper limit of confidence interval could not be estimated due to insufficient events. | NA [7.14 to NA] — Here, NA means median and upper limit of confidence interval could not be estimated due to insufficient events. | NA [NA to NA] — Here, NA means median and confidence interval could not be estimated due to insufficient events. | 39.07 [13.14 to 65.00] | 27.86 [NA to NA] — Here, NA means lower and upper limit of confidence interval could not be estimated due to insufficient events.

14. Secondary Outcome: Parts B, and C: Immune DOR (iDOR) Based on iRECIST
Description: iDOR was defined as the time from the first documentation of response (iCR or iPR) to the first documentation of objective tumor progression (immune confirmed progressive disease [iCPD]) or death due to any cause based on iRECIST.
Time Frame: From first dose of study drug up to 40.3 months for Part B; up to 50.5 months for Part C
Population: as for outcome 12
Arm/Group | Part B, Dose Expansion, Melanoma: Nemvaleukin Alfa 6 mcg/kg | Part B, Dose Expansion, RCC: Nemvaleukin Alfa 6 mcg/kg | Part C, Combination Therapy, Safety Run-in: Nemvaleukin Alfa 1 mcg/kg | Part C, Combination Therapy, Cohort 1 +Safety Run-in: Nemvaleukin Alfa 3 mcg/kg+Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 2: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 3: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Rollover, Cohort 4: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 5: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 6: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 7: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

15. Secondary Outcome: Part B and Part C Cohorts C5, C6, C7: Durable Response Rate (DRR) Based on RECIST v.1.1
Description: DRR was defined as the percentage of participants with an objective response (complete or partial response per RECIST 1.1) lasting continuously for 6 months and starting any time within 12 months of initiating the study drug.
Time Frame: From first dose of study drug up to 40.3 months for Part B; up to 50.5 months for Part C
Population: As pre-specified in statistical analysis plan, this outcome measure of DRR was not summarized and hence, no data was reported in this outcome measure.
Arm/Group | Part B, Dose Expansion, Melanoma: Nemvaleukin Alfa 6 mcg/kg | Part B, Dose Expansion, RCC: Nemvaleukin Alfa 6 mcg/kg | Part C, Combination Therapy, Cohort 5: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 6: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 7: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

16. Secondary Outcome: Part B and Part C Cohorts C5, C6, C7: Immune DRR (iDRR) Based on iRECIST
Description: iDRR was defined as the percentage of participants with an objective response (complete or partial response per iRECIST) lasting continuously for 6 months and starting any time within 12 months of initiating the study drug.
Time Frame: From first dose of study drug up to 40.3 months for Part B; up to 50.5 months for Part C
Population: as for outcome 12
Arm/Group | Part B, Dose Expansion, Melanoma: Nemvaleukin Alfa 6 mcg/kg | Part B, Dose Expansion, RCC: Nemvaleukin Alfa 6 mcg/kg | Part C, Combination Therapy, Cohort 5: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 6: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 7: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

17. Secondary Outcome: Part B and Part C Cohorts C5, C6, C7: Progression-free Survival (PFS) Based on RECIST v.1.1
Description: Progression-free survival was defined as the time from the first dose of nemvaleukin to the first documentation of objective tumor progression or death due to any cause. PD: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this included the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: From first dose of study drug up to the first documentation of objective tumor progression or death due to any cause (up to 40.3 months for Part B and up to 50.5 months for Part C)
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Part B, Dose Expansion, Melanoma: Nemvaleukin Alfa 6 mcg/kg | Part B, Dose Expansion, RCC: Nemvaleukin Alfa 6 mcg/kg | Part C, Combination Therapy, Cohort 5: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 6: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 7: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg
Number analyzed (Participants) | 46 | 22 | 3 | 18 | 2
weeks | 16.14 [10.57 to 17.14] | 12.43 [4.43 to 22.57] | NA [10.29 to NA] — Here, NA means median and upper limit of confidence interval could not be estimated due to insufficient events. | 18.64 [6.14 to 27.14] | 35.57 [18.71 to 52.43]

18. Secondary Outcome: Part B and Part C Cohorts C5, C6, C7: Immune PFS (iPFS)
Description: iPFS was defined as the time from the first dose of study medication to the first documentation of objective tumor progression based on iRECIST (immune confirmed progressive disease [iCPD]) or death due to any cause.
Time Frame: From first dose of study drug up to 40.3 months for Part B; up to 50.5 months for Part C
Population: as for outcome 12
Arm/Group | Part B, Dose Expansion, Melanoma: Nemvaleukin Alfa 6 mcg/kg | Part B, Dose Expansion, RCC: Nemvaleukin Alfa 6 mcg/kg | Part C, Combination Therapy, Cohort 5: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 6: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 7: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

19. Secondary Outcome: Parts A, B and C: Maximum Cell Count of Whole Blood FoxP3+ T Cells (Tregs), Total Cluster of Differentiation (CD)8+ T Cells and Natural Killer (NK) Cells
Time Frame: Cycle 1 Day 1 (Cycle 1 length = 14 days for Part A and 21 days for Part B and C)
Population: The pharmacodynamic (PD) population consisted of all participants who received at least 1 dose of nemvaleukin alfa and had at least one available postbaseline PD measurement. Here, "overall number of participants analyzed" signifies participants who were evaluable for this outcome measure and "number analyzed" signifies participants who were evaluable at specified timepoints.
Measure: Mean (Standard Deviation); unit: cells per microliters (cells/mcL)
Arm/Group | Part A, Dose Escalation: Nemvaleukin Alfa 0.1 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 0.3 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 1 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 3 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 6 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 8 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 10 mcg/kg | Part B, Dose Expansion, Melanoma: Nemvaleukin Alfa 6 mcg/kg | Part B, Dose Expansion, RCC: Nemvaleukin Alfa 6 mcg/kg | Part C, Combination Therapy, Safety Run-in: Nemvaleukin Alfa 1 mcg/kg | Part C, Combination Therapy, Safety Run-in: Nemvaleukin Alfa 3 mcg/kg | Part C, Combination Therapy, Cohort 1: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 2: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 3: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Rollover, Cohort 4: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 5: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 6: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 7: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg
Number analyzed (Participants) | 5 | 4 | 7 | 8 | 12 | 3 | 7 | 27 | 47 | 3 | 6 | 36 | 25 | 26 | 39 | 3 | 21 | 2
cells per microliters (cells/mcL)
  Whole Blood FoxP3+ T Cells (Tregs): number analyzed (Participants) | 5 | 4 | 7 | 8 | 12 | 3 | 7 | 27 | 47 | 3 | 6 | 36 | 25 | 26 | 39 | 3 | 21 | 1
  Whole Blood FoxP3+ T Cells (Tregs) | 32.0 (11.3) | 50.5 (53.7) | 56.6 (22.3) | 46.3 (21.8) | 43.3 (28.2) | 57.4 (14.4) | 51.3 (36.0) | 40.3 (23.5) | 47.9 (24.0) | 27.4 (7.31) | 50.9 (23.9) | 42.6 (28.3) | 37.8 (24.5) | 41.6 (27.7) | 44.3 (22.5) | 51.1 (9.85) | 52.6 (31.3) | 33.1 (NA) — Standard Deviation could not be calculated for 1 participant.
  Total CD8+ T Cells | 247 (107) | 204 (89.2) | 262 (64.2) | 466 (255) | 610 (570) | 704 (559) | 703 (502) | 1392 (1053) | 773 (422) | 262 (186) | 551 (433) | 562 (373) | 533 (328) | 688 (384) | 718 (567) | 924 (638) | 762 (538) | 445 (349)
  NK Cells | 197 (61.4) | 343 (20.6) | 467 (313) | 685 (307) | 1053 (660) | 978 (400) | 1038 (1028) | 1279 (642) | 1470 (873) | 531 (296) | 804 (196) | 771 (503) | 760 (458) | 813 (436) | 889 (438) | 1081 (787) | 1064 (445) | 1298 (334)

20. Secondary Outcome: Parts A, B and C: Maximum Cell Count of Interferon-gamma (INF-γ) and Interleukin 6 (IL-6)
Time Frame: Cycle 1 Days 1 and 5; Cycle 2 Days 1 and 5 (Cycle 1 length = 14 days for Part A and 21 days for Part B and C; Cycle 2 length= 21 days for all parts)
Population: The PD population consisted of all participants who received at least 1 dose of nemvaleukin alfa and had at least one available postbaseline PD measurement. Here, "overall number of participants analyzed" signifies participants who were evaluable for this outcome measure and "number analyzed" signifies participants who were evaluable at specified timepoints.
Measure: Mean (Standard Deviation); unit: nanogram per liter (ng/L)
Arm/Group | Part A, Dose Escalation: Nemvaleukin Alfa 0.1 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 0.3 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 1 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 3 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 6 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 8 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 10 mcg/kg | Part B, Dose Expansion, Melanoma: Nemvaleukin Alfa 6 mcg/kg | Part B, Dose Expansion, RCC: Nemvaleukin Alfa 6 mcg/kg | Part C, Combination Therapy, Safety Run-in: Nemvaleukin Alfa 1 mcg/kg | Part C, Combination Therapy, Safety Run-in: Nemvaleukin Alfa 3 mcg/kg | Part C, Combination Therapy, Cohort 1: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 2: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 3: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Rollover, Cohort 4: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 5: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 6: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 7: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg
Number analyzed (Participants) | 5 | 4 | 7 | 8 | 10 | 2 | 7 | 34 | 15 | 3 | 6 | 31 | 17 | 20 | 21 | 2 | 18 | 2
nanogram per liter (ng/L)
  INF-γ: Cycle 1 Day 1: number analyzed (Participants) | 5 | 4 | 7 | 8 | 10 | 1 | 7 | 12 | 15 | 0 | 2 | 29 | 4 | 3 | 21 | 1 | 5 | 0
  INF-γ: Cycle 1 Day 1 | 23.0 (10.3) | 19.8 (10.4) | 14.9 (6.10) | 31.3 (12.7) | 108 (130) | 26.4 (NA) — Standard Deviation could not be calculated for a single participant. | 18.0 (NA) — Standard Deviation could not be calculated for a single participant. | 34.7 (22.7) | 18.6 (4.19) |  | 23.3 (7.40) | 77.0 (106) | 34.5 (15.6) | 18.9 (3.71) | 84.4 (87.8) | 68.3 (NA) — Standard Deviation could not be calculated for a single participant. | 31.7 (24.2) |
  INF-γ: Cycle 1 Day 5: number analyzed (Participants) | 5 | 4 | 5 | 7 | 8 | 2 | 4 | 34 | 13 | 0 | 4 | 29 | 14 | 17 | 17 | 2 | 17 | 2
  INF-γ: Cycle 1 Day 5 | 24.7 (10.8) | 29.1 (10.7) | 13.8 (7.71) | 173 (199) | 129 (84.1) | 585 (313) | 335 (74.3) | 209 (191) | 162 (183) |  | 48.2 (30.3) | 92.6 (86.4) | 94.3 (103) | 70.9 (54.7) | 64.4 (61.5) | 390 (530) | 279 (526) | 87.7 (42.1)
  INF-γ: Cycle 2 Day 1: number analyzed (Participants) | 4 | 4 | 5 | 5 | 1 | 2 | 1 | 16 | 4 | 0 | 1 | 7 | 5 | 4 | 4 | 1 | 3 | 0
  INF-γ: Cycle 2 Day 1 | 28.0 (24.1) | 18.3 (3.70) | 12.2 (4.56) | 43.3 (28.4) | 33.9 (NA) — Standard Deviation could not be calculated for a single participant. | 19.8 (4.81) | 15.7 (NA) — Standard Deviation could not be calculated for a single participant. | 43.3 (41.9) | 50.4 (22.7) |  | 15.4 (NA) — Standard Deviation could not be calculated for a single participant. | 70.9 (102) | 21.1 (6.39) | 19.7 (3.87) | 62.4 (20.7) | 43.5 (NA) — Standard Deviation could not be calculated for a single participant. | 25.8 (1.04) |
  INF-γ: Cycle 2 Day 5: number analyzed (Participants) | 3 | 4 | 6 | 5 | 6 | 2 | 3 | 33 | 10 | 0 | 4 | 20 | 10 | 17 | 21 | 2 | 12 | 2
  INF-γ: Cycle 2 Day 5 | 31.2 (19.2) | 24.3 (10.8) | 16.3 (8.03) | 53.2 (15.3) | 45.1 (28.5) | 171 (78.4) | 84.8 (58.6) | 141 (139) | 120 (178) |  | 60.3 (19.5) | 73.3 (77.7) | 47.7 (43.5) | 38.5 (22.2) | 54.0 (36.1) | 326 (124) | 101 (71.0) | 41.9 (1.42)
  IL-6: Cycle 1 Day 1: number analyzed (Participants) | 5 | 3 | 7 | 8 | 10 | 2 | 6 | 29 | 13 | 0 | 5 | 29 | 16 | 18 | 14 | 2 | 15 | 0
  IL-6: Cycle 1 Day 1 | 104 (61.8) | 118 (33.0) | 169 (280) | 938 (845) | 254 (177) | 148 (14.6) | 1826 (3474) | 323 (630) | 211 (143) |  | 506 (137) | 667 (1020) | 274 (234) | 306 (181) | 706 (1757) | 200 (101) | 757 (2165) |
  IL-6: Cycle 1 Day 5: number analyzed (Participants) | 5 | 4 | 7 | 7 | 9 | 2 | 4 | 33 | 15 | 1 | 5 | 31 | 17 | 20 | 16 | 2 | 18 | 2
  IL-6: Cycle 1 Day 5 | 116 (121) | 113 (51.9) | 223 (229) | 2022 (1491) | 802 (797) | 677 (751) | 5240 (5279) | 699 (538) | 723 (1077) | 151 (NA) — Standard Deviation could not be calculated for a single participant. | 524 (180) | 1269 (1807) | 513 (585) | 527 (538) | 273 (244) | 1049 (1288) | 635 (500) | 232 (13.8)
  IL-6: Cycle 2 Day 1: number analyzed (Participants) | 5 | 4 | 7 | 6 | 6 | 2 | 4 | 31 | 12 | 1 | 6 | 23 | 15 | 12 | 11 | 2 | 12 | 0
  IL-6: Cycle 2 Day 1 | 41.9 (14.7) | 106 (76.4) | 191 (240) | 883 (570) | 351 (448) | 169 (18.1) | 519 (475) | 311 (447) | 254 (151) | 95.7 (NA) — Standard Deviation could not be calculated for a single participant. | 254 (99.4) | 669 (1075) | 276 (249) | 372 (279) | 282 (176) | 718 (649) | 264 (379) |
  IL-6: Cycle 2 Day 5: number analyzed (Participants) | 3 | 4 | 7 | 5 | 5 | 2 | 3 | 30 | 10 | 3 | 6 | 21 | 17 | 12 | 15 | 2 | 12 | 2
  IL-6: Cycle 2 Day 5 | 56.2 (19.1) | 95.2 (45.3) | 125 (89.3) | 1145 (700) | 399 (243) | 252 (124) | 1372 (1841) | 341 (252) | 318 (174) | 116 (33.0) | 425 (339) | 929 (1962) | 290 (296) | 269 (155) | 269 (174) | 165 (98.6) | 267 (172) | 123 (19.0)

ADVERSE EVENTS:
Time Frame: From first dose of study drug until 30 days after last dose (up to 10 months for Part A; up to 41.3 months for Part B; up to 51.5 months for Part C)
Arm/Group | Part A, Dose Escalation: Nemvaleukin Alfa 0.1 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 0.3 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 1 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 3 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 6 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 8 mcg/kg | Part A, Dose Escalation: Nemvaleukin Alfa 10 mcg/kg | Part B, Dose Expansion, Melanoma: Nemvaleukin Alfa 6 mcg/kg | Part B, Dose Expansion, RCC: Nemvaleukin Alfa 6 mcg/kg | Part C, Combination Therapy, Safety Run-in: Nemvaleukin Alfa 1 mcg/kg | Part C, Combination Therapy, Cohort 1 +Safety Run-in: Nemvaleukin Alfa 3 mcg/kg +Pembrolizumab 200mg | Part C, Combination Therapy, Cohort 2: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 3: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Rollover, Cohort 4: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 5: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 6: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg | Part C, Combination Therapy, Cohort 7: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4 | 0/7 | 0/8 | 1/12 | 0/3 | 3/7 | 7/47 | 7/27 | 0/3 | 7/42 | 7/26 | 8/26 | 8/43 | 1/3 | 8/21 | 1/2
Serious Adverse Events (participants affected / at risk) | 2/5 | 0/4 | 2/7 | 3/8 | 5/12 | 0/3 | 5/7 | 11/47 | 12/27 | 0/3 | 19/42 | 10/26 | 11/26 | 14/43 | 2/3 | 12/21 | 2/2
Other Adverse Events (participants affected / at risk) | 5/5 | 4/4 | 7/7 | 8/8 | 12/12 | 3/3 | 7/7 | 46/47 | 27/27 | 3/3 | 42/42 | 26/26 | 25/26 | 38/43 | 3/3 | 21/21 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A, Dose Escalation: Nemvaleukin Alfa 0.1 mcg/kg (N=5) | Part A, Dose Escalation: Nemvaleukin Alfa 0.3 mcg/kg (N=4) | Part A, Dose Escalation: Nemvaleukin Alfa 1 mcg/kg (N=7) | Part A, Dose Escalation: Nemvaleukin Alfa 3 mcg/kg (N=8) | Part A, Dose Escalation: Nemvaleukin Alfa 6 mcg/kg (N=12) | Part A, Dose Escalation: Nemvaleukin Alfa 8 mcg/kg (N=3) | Part A, Dose Escalation: Nemvaleukin Alfa 10 mcg/kg (N=7) | Part B, Dose Expansion, Melanoma: Nemvaleukin Alfa 6 mcg/kg (N=47) | Part B, Dose Expansion, RCC: Nemvaleukin Alfa 6 mcg/kg (N=27) | Part C, Combination Therapy, Safety Run-in: Nemvaleukin Alfa 1 mcg/kg (N=3) | Part C, Combination Therapy, Cohort 1 +Safety Run-in: Nemvaleukin Alfa 3 mcg/kg +Pembrolizumab 200mg (N=42) | Part C, Combination Therapy, Cohort 2: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg (N=26) | Part C, Combination Therapy, Cohort 3: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg (N=26) | Part C, Combination Therapy, Rollover, Cohort 4: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg (N=43) | Part C, Combination Therapy, Cohort 5: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg (N=3) | Part C, Combination Therapy, Cohort 6: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg (N=21) | Part C, Combination Therapy, Cohort 7: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg (N=2)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (5) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Extravasation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram T wave abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Troponin I increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iritis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitritis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess neck (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthritis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peritoneal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular device infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 4 (6) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myelopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Starvation (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Stomal hernia (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embolism arterial (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection enterococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A, Dose Escalation: Nemvaleukin Alfa 0.1 mcg/kg (N=5) | Part A, Dose Escalation: Nemvaleukin Alfa 0.3 mcg/kg (N=4) | Part A, Dose Escalation: Nemvaleukin Alfa 1 mcg/kg (N=7) | Part A, Dose Escalation: Nemvaleukin Alfa 3 mcg/kg (N=8) | Part A, Dose Escalation: Nemvaleukin Alfa 6 mcg/kg (N=12) | Part A, Dose Escalation: Nemvaleukin Alfa 8 mcg/kg (N=3) | Part A, Dose Escalation: Nemvaleukin Alfa 10 mcg/kg (N=7) | Part B, Dose Expansion, Melanoma: Nemvaleukin Alfa 6 mcg/kg (N=47) | Part B, Dose Expansion, RCC: Nemvaleukin Alfa 6 mcg/kg (N=27) | Part C, Combination Therapy, Safety Run-in: Nemvaleukin Alfa 1 mcg/kg (N=3) | Part C, Combination Therapy, Cohort 1 +Safety Run-in: Nemvaleukin Alfa 3 mcg/kg +Pembrolizumab 200mg (N=42) | Part C, Combination Therapy, Cohort 2: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg (N=26) | Part C, Combination Therapy, Cohort 3: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg (N=26) | Part C, Combination Therapy, Rollover, Cohort 4: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg (N=43) | Part C, Combination Therapy, Cohort 5: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg (N=3) | Part C, Combination Therapy, Cohort 6: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg (N=21) | Part C, Combination Therapy, Cohort 7: Nemvaleukin Alfa 6 mcg/kg + Pembrolizumab 200 mg (N=2)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 5 (8) | 8 (24) | 12 (59) | 2 (10) | 3 (7) | 33 (104) | 17 (27) | 1 (1) | 30 (148) | 17 (80) | 16 (45) | 7 (33) | 2 (7) | 10 (37) | 2 (29)
Chills (General disorders) | 0 (0) | 2 (8) | 5 (16) | 8 (29) | 11 (52) | 3 (32) | 2 (2) | 21 (226) | 14 (47) | 1 (3) | 32 (171) | 16 (62) | 18 (95) | 9 (129) | 3 (7) | 13 (65) | 2 (42)
Fatigue (General disorders) | 4 (6) | 1 (1) | 2 (2) | 3 (4) | 4 (5) | 2 (9) | 3 (7) | 11 (28) | 8 (14) | 1 (2) | 19 (33) | 8 (8) | 11 (39) | 9 (28) | 3 (6) | 6 (11) | 2 (18)
Oedema peripheral (General disorders) | 1 (2) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 1 (2) | 5 (6) | 1 (1) | 2 (7) | 8 (13) | 3 (3) | 5 (10) | 1 (1) | 2 (3) | 2 (2) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 1 (2) | 1 (1) | 2 (4) | 2 (2) | 2 (5) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (10) | 3 (3) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (4) | 2 (2) | 2 (2) | 4 (10) | 5 (9) | 3 (14) | 0 (0) | 13 (29) | 3 (3) | 1 (1) | 15 (27) | 8 (13) | 10 (23) | 4 (49) | 2 (2) | 8 (13) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (3) | 1 (1) | 1 (4) | 4 (8) | 5 (13) | 3 (6) | 0 (0) | 24 (90) | 8 (10) | 0 (0) | 21 (45) | 13 (22) | 9 (36) | 8 (64) | 1 (1) | 12 (29) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (5) | 4 (4) | 1 (1) | 3 (8) | 1 (1) | 6 (12) | 3 (3) | 0 (0) | 15 (20) | 5 (6) | 5 (6) | 3 (6) | 0 (0) | 5 (5) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (5) | 1 (1) | 3 (9) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 11 (12) | 3 (4) | 5 (6) | 4 (6) | 0 (0) | 2 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2) | 2 (3) | 1 (1) | 1 (1) | 1 (1) | 6 (26) | 3 (3) | 1 (1) | 10 (15) | 5 (5) | 8 (13) | 11 (20) | 0 (0) | 4 (6) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (2) | 0 (0) | 3 (3) | 7 (16) | 1 (1) | 4 (7) | 20 (65) | 5 (8) | 0 (0) | 18 (67) | 4 (4) | 6 (11) | 4 (7) | 0 (0) | 6 (54) | 1 (4)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (6) | 2 (5) | 2 (6) | 0 (0) | 4 (15) | 3 (3) | 0 (0) | 4 (5) | 3 (6) | 6 (18) | 1 (6) | 1 (2) | 4 (7) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 3 (4) | 4 (4) | 0 (0) | 1 (2) | 0 (0) | 2 (5) | 6 (8) | 0 (0) | 8 (17) | 1 (2) | 4 (5) | 4 (6) | 0 (0) | 3 (3) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 1 (1) | 2 (4) | 17 (27) | 6 (8) | 0 (0) | 4 (11) | 3 (5) | 8 (17) | 5 (27) | 1 (1) | 5 (9) | 1 (3)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 3 (6) | 18 (27) | 7 (10) | 0 (0) | 6 (9) | 3 (6) | 8 (19) | 5 (24) | 1 (1) | 3 (5) | 1 (2)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 4 (4) | 2 (2) | 0 (0) | 6 (20) | 0 (0) | 4 (7) | 2 (2) | 0 (0) | 5 (14) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (28) | 2 (2) | 3 (15) | 3 (8) | 0 (0) | 4 (24) | 1 (3)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 2 (3) | 4 (4) | 1 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 3 (7) | 2 (2) | 1 (1) | 7 (51) | 3 (4) | 4 (26) | 0 (0) | 0 (0) | 8 (72) | 1 (10)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 2 (4) | 11 (21) | 7 (7) | 0 (0) | 13 (15) | 3 (3) | 13 (15) | 2 (5) | 1 (2) | 6 (6) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 1 (4) | 0 (0) | 4 (7) | 2 (2) | 0 (0) | 8 (24) | 8 (10) | 5 (7) | 2 (3) | 0 (0) | 4 (5) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 4 (6) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1) | 3 (8) | 2 (2) | 1 (1) | 2 (2) | 5 (6) | 8 (9) | 1 (1) | 8 (10) | 4 (5) | 6 (14) | 0 (0) | 1 (1) | 11 (40) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 6 (13) | 3 (4) | 0 (0) | 5 (5) | 2 (5) | 2 (3) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 3 (3) | 2 (2) | 1 (1) | 13 (26) | 6 (40) | 0 (0) | 10 (19) | 8 (9) | 9 (32) | 8 (15) | 2 (2) | 4 (7) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (2) | 2 (3) | 2 (4) | 0 (0) | 1 (2) | 1 (1) | 6 (12) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 6 (8) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 1 (1) | 2 (2) | 2 (3) | 1 (3) | 0 (0) | 7 (19) | 3 (8) | 1 (1) | 7 (9) | 2 (2) | 4 (6) | 4 (7) | 0 (0) | 4 (10) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (2) | 0 (0) | 5 (18) | 3 (3) | 0 (0) | 6 (13) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 1 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 3 (14) | 1 (1) | 0 (0) | 7 (9) | 0 (0) | 2 (6) | 3 (4) | 0 (0) | 2 (11) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 7 (7) | 2 (2) | 0 (0) | 6 (7) | 3 (3) | 7 (26) | 7 (15) | 1 (1) | 4 (4) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 4 (23) | 0 (0) | 0 (0) | 7 (10) | 5 (18) | 0 (0) | 16 (59) | 2 (2) | 6 (24) | 4 (6) | 0 (0) | 6 (20) | 1 (2)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (7) | 0 (0) | 1 (2) | 0 (0) | 4 (5) | 2 (4) | 0 (0) | 3 (3) | 3 (8) | 3 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 4 (10) | 4 (7) | 0 (0) | 6 (7) | 1 (1) | 3 (3) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (9) | 2 (7) | 0 (0) | 3 (6) | 5 (6) | 6 (8) | 4 (5) | 0 (0) | 3 (5) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 1 (4) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 31 (152) | 11 (49) | 0 (0) | 8 (58) | 4 (5) | 10 (68) | 15 (83) | 2 (15) | 7 (33) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 3 (3) | 3 (12) | 1 (1) | 2 (5) | 5 (7) | 15 (38) | 8 (17) | 2 (2) | 13 (35) | 5 (9) | 11 (32) | 13 (34) | 1 (1) | 9 (38) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 5 (8) | 3 (4) | 0 (0) | 10 (42) | 1 (1) | 3 (6) | 2 (2) | 2 (2) | 2 (7) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (9) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 0 (0) | 5 (6) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 5 (17) | 0 (0) | 4 (18) | 4 (19) | 2 (2) | 1 (1) | 1 (3) | 2 (8) | 0 (0)
Blood pressure (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (25) | 6 (11) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (9) | 2 (3) | 1 (1) | 6 (73) | 1 (2) | 4 (53) | 0 (0) | 1 (1) | 6 (35) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 1 (1) | 0 (0) | 4 (6) | 2 (2) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (7) | 0 (0) | 4 (5) | 4 (5) | 2 (2) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 2 (6) | 0 (0) | 2 (7) | 1 (1) | 3 (3) | 3 (7) | 0 (0) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 4 (12) | 1 (3)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 1 (1) | 3 (5) | 3 (4) | 0 (0) | 2 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (15) | 0 (0) | 2 (5) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (7) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 5 (5) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (5) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 2 (4) | 1 (1) | 1 (1) | 0 (0) | 2 (10) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 1 (1) | 2 (5) | 1 (1) | 0 (0) | 2 (5) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (4) | 1 (1) | 3 (9) | 1 (3) | 3 (4) | 5 (8) | 0 (0) | 4 (6) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2022-09-08): https://cdn.clinicaltrials.gov/large-docs/95/NCT02799095/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-03): https://cdn.clinicaltrials.gov/large-docs/95/NCT02799095/SAP_001.pdf